CLINICAL TRIAL: NCT01193127
Title: Safety and Efficacy of OMS302 in Subjects Undergoing Unilateral Cataract Extraction With Lens Replacement (CELR)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Omeros Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: C09-001
Record Dates: First submitted 2010-08-23; First posted 2010-09-01 (Estimated); Results first posted 2014-08-28 (Estimated); Last update posted 2014-08-28 (Estimated); Status verified 2014-08

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract | interventions — Solutions

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- OMS302 Solution (Experimental): OMS302 Solution
  Interventions: Drug: OMS302 Solution
- OMS302 Mydriatic Solution (Experimental): OMS302 Mydriatic Solution
  Interventions: Drug: OMS302 Mydriatic Solution
- OMS302 Anti-inflammatory Solution (Experimental): OMS302 Anti-inflammatory Solution
  Interventions: Drug: OMS302 Anti-inflammatory Solution
- Balanced Salt Solution (BSS) Solution (Placebo Comparator): Balanced Salt Solution (BSS) Solution
  Interventions: Drug: Balanced Salt Solution (BSS) Solution

INTERVENTIONS:
Drug: OMS302 Solution
  Arms: OMS302 Solution
Drug: OMS302 Mydriatic Solution
  Arms: OMS302 Mydriatic Solution
Drug: OMS302 Anti-inflammatory Solution
  Arms: OMS302 Anti-inflammatory Solution
Drug: Balanced Salt Solution (BSS) Solution
  Arms: Balanced Salt Solution (BSS) Solution

SUMMARY:
The purpose of this study is to determine whether the use of OMS302 (the study drug) in individuals undergoing Cataract Extraction with Lens Replacement (CELR) surgery is safe and effective at maintaining an adequately dilated pupil during surgery and reducing post-operative symptoms of discomfort (such as eye pain and irritation).

ELIGIBILITY:
Inclusion Criteria:

* Competent and willing to voluntarily provide informed consent
* 18 years of age or older
* In good general health needing to undergo cataract extraction with lens replacement surgery in one eye, under topical anesthesia
* Other inclusion criteria to be evaluated by the investigator

Exclusion Criteria:

* No allergies to the medications and/or the active ingredients of any of the study medications
* No medications with the same activities as the of the active ingredients in OMS302 for defined time intervals prior to and after surgery
* No other significant eye injuries, eye conditions or general medical conditions likely to interfere with the evaluation of the study medication
* Other exclusion criteria to be evaluated by the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 223 (Actual)
Dates: Start 2010-07; Primary Completion 2011-01 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (24):
- United States (24):
  - Chandler, Arizona
  - Glendale, Arizona
  - Little Rock, Arkansas
  - Los Angeles, California
  - Parker, Colorado
  - Largo, Florida
  - North Fort Myers, Florida
  - Panama City, Florida
  - Tamarac, Florida
  - Gurnee, Illinois
  - Gretna, Louisiana
  - Kansas City, Missouri
  - St Louis, Missouri
  - Omaha, Nebraska
  - Las Vegas, Nevada
  - Albuquerque, New Mexico
  - Rockville Centre, New York
  - Bala-Cynwyd, Pennsylvania
  - Goodlettsville, Tennessee
  - Austin, Texas
  - Houston, Texas
  - Nacogdoches, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah

RESULTS

PARTICIPANT FLOW:
Groups:
- Balanced Salt Solution (BSS): Balanced Salt Solution (BSS)
  Balanced Salt Solution (BSS)
- OMS302 Mydriatic Solution (PE): OMS302 Mydriatic Solution
  OMS302 Mydriatic Solution
- OMS302 Anti-inflammatory Solution (KE): OMS302 Anti-inflammatory Solution
  OMS302 Anti-inflammatory Solution
Period: Randomized
Arm/Group | Balanced Salt Solution (BSS) | OMS302 Mydriatic Solution (PE) | OMS302 Anti-inflammatory Solution (KE) | OMS302 Solution
Started | 57 | 54 | 55 | 57
Completed | 57 | 54 | 55 | 56
Not Completed | 0 | 0 | 0 | 1
Not completed — Surgery Cancelled | 0 | 0 | 0 | 1
Period: Treated
Arm/Group | Balanced Salt Solution (BSS) | OMS302 Mydriatic Solution (PE) | OMS302 Anti-inflammatory Solution (KE) | OMS302 Solution
Started | 57 | 54 | 55 | 56
Completed | 57 | 54 | 55 | 55
Not Completed | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Balanced Salt Solution (BSS) | OMS302 Mydriatic Solution (PE) | OMS302 Anti-inflammatory Solution (KE) | OMS302 Solution | Total
Number analyzed (Participants) | 57 | 54 | 55 | 56 | 222
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.5 (9.6) | 67.6 (10.6) | 66.8 (8.6) | 66.4 (11.2) | 67.3 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 34 | 33 | 37 | 137
  Male | 24 | 20 | 22 | 19 | 85

OUTCOME MEASURES:

1. Primary Outcome: Pupil Diameter (mm) During Surgery
Description: Pupil diameter from surgical baseline (immediately prior to surgical incision) to the end of the surgical procedure (wound closure) was summarized using descriptive statistics by treatment group and time point. Repeated measures analyses of variance were used to test for differences in the maintenance of mydriasis. The repeated measures model included change from baseline pupil diameter as the response variable and treatment (OMS302, ketorolac tromethamine, and vehicle), time point (as a categorical variable) and the stratification factor lens opacities classification system II (LOCS II) grade as predictor variables. A generalized estimating equation (GEE) approach with an AR(1) working-correlation structure was used.
Time Frame: During surgery (immediately prior to surgical incision to wound closure)
Population: Subjects with interpretable video recordings obtained during surgery.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Balanced Salt Solution (BSS) | OMS302 Mydriatic Solution (PE) | OMS302 Anti-inflammatory Solution (KE) | OMS302 Solution
Number analyzed (Participants) | 53 | 49 | 52 | 49
mm
  Baseline; n = 53, 49, 52, 49 | 8.0 (2.0) | 8.0 (1.8) | 8.1 (1.6) | 9.0 (2.9)
  1 minute; n = 53, 48, 52, 48 | 8.2 (2.1) | 8.3 (1.9) | 8.3 (1.6) | 9.4 (3.1)
  2 minutes; n = 53, 49, 52, 49 | 8.0 (2.0) | 8.3 (1.7) | 8.2 (1.8) | 9.2 (3.2)
  3 minutes; n = 53, 49, 52, 49 | 7.9 (2.2) | 8.4 (1.8) | 8.1 (1.7) | 9.2 (3.1)
  4 minutes; n = 52, 49, 52, 49 | 7.6 (2.0) | 8.4 (1.8) | 7.9 (1.8) | 9.4 (3.1)
  5 minutes; n = 52, 49, 51, 48 | 7.5 (2.3) | 8.2 (1.9) | 7.9 (1.9) | 9.1 (2.8)
  6 minutes; n = 51, 45, 50, 48 | 7.4 (2.6) | 8.1 (2.0) | 7.7 (1.8) | 9.1 (3.1)
  7 minutes; n = 45, 37, 44, 43 | 7.1 (2.7) | 8.0 (2.3) | 7.2 (2.0) | 9.0 (3.1)
  8 minutes; n = 34, 28, 40, 36 | 7.1 (2.7) | 7.8 (2.5) | 7.1 (2.1) | 8.7 (3.0)
  9 minutes; n = 27, 25, 32, 32 | 7.3 (3.0) | 8.1 (2.6) | 7.0 (1.9) | 8.9 (3.0)
  10 minutes; n = 26, 19, 25, 28 | 7.1 (2.5) | 8.3 (2.8) | 7.0 (1.5) | 8.8 (3.2)
  11 minutes; n = 24, 18, 22, 27 | 7.0 (2.9) | 8.3 (2.7) | 7.1 (1.4) | 8.8 (3.2)
  12 minutes; n = 22, 17, 20, 23 | 6.9 (3.0) | 8.0 (2.7) | 7.0 (1.1) | 9.2 (3.8)
  13 minutes; n = 14, 13, 16, 17 | 6.2 (1.6) | 8.0 (2.9) | 6.8 (1.4) | 8.7 (3.3)
  14 minutes; n = 10, 8, 13, 10 | 6.3 (1.8) | 7.7 (2.8) | 6.5 (1.4) | 9.5 (3.0)
  15 minutes; n = 8, 7, 8, 9 | 6.1 (1.6) | 7.9 (2.7) | 6.9 (2.1) | 9.9 (3.7)
  16 minutes; n = 7, 6, 7, 6 | 5.8 (1.9) | 8.4 (3.0) | 6.7 (1.6) | 10.4 (4.8)
  17 minutes; n = 7, 5, 6, 5 | 5.6 (1.8) | 7.2 (1.4) | 6.8 (1.7) | 12.0 (5.1)
  18 minutes; n = 6, 3, 5, 5 | 5.4 (1.6) | 7.9 (0.9) | 6.8 (3.1) | 12.0 (5.6)
  19 minutes; n = 3, 3, 4, 5 | 5.2 (2.1) | 7.8 (1.0) | 6.7 (3.9) | 11.5 (5.0)
  20 minutes; n = 2, 2, 2, 3 | 5.2 (3.2) | 8.1 (1.4) | 5.2 (0.9) | 12.4 (6.3)
  21 minutes; n = 2, 2, 0, 3 | 4.9 (3.3) | 8.0 (1.5) | NA (NA) — No subjects in this treatment group continuing surgery past this time point. | 12.0 (5.8)
  22 minutes; n = 1, 2, 0, 2 | 2.3 (0) | 7.5 (1.5) | NA (NA) — No subjects in this treatment group continuing surgery past this time point. | 14.6 (7.6)
  23 minutes; n = 1, 1, 0, 2 | 3.0 (0) | 6.6 (0) | NA (NA) — No subjects in this treatment group continuing surgery past this time point. | 14.6 (7.1)
  24 minutes; n = 1, 1, 0, 2 | 4.2 (0) | 7.1 (0) | NA (NA) — No subjects in this treatment group continuing surgery past this time point. | 13.0 (5.7)
  25 minutes; n = 1, 1, 0, 2 | 2.6 (0) | 6.4 (0) | NA (NA) — No subjects in this treatment group continuing surgery past this time point. | 13.9 (5.9)
  26 minutes; n = 1, 0, 0, 1 | 3.1 (0) | NA (NA) — No subjects in this treatment group continuing surgery past this time point. | NA (NA) — No subjects in this treatment group continuing surgery past this time point. | 17.2 (0)
  27 minutes; n = 1, 0, 0, 1 | 3.3 (0) | NA (NA) — No subjects in this treatment group continuing surgery past this time point. | NA (NA) — No subjects in this treatment group continuing surgery past this time point. | 17.4 (0)
  28 minutes; n = 1, 0, 0, 1 | 3.6 (0) | NA (NA) — No subjects in this treatment group continuing surgery past this time point. | NA (NA) — No subjects in this treatment group continuing surgery past this time point. | 17.1 (0)
  29 minutes; n = 1, 0, 0, 1 | 3.4 (0) | NA (NA) — No subjects in this treatment group continuing surgery past this time point. | NA (NA) — No subjects in this treatment group continuing surgery past this time point. | 18.7 (0)
  30 minutes; n = 1, 0, 0, 0 | 4.1 (0) | NA (NA) — No subjects in this treatment group continuing surgery past this time point. | NA (NA) — No subjects in this treatment group continuing surgery past this time point. | NA (NA) — No subjects in this treatment group continuing surgery past this time point.
  31 minutes; n = 1, 0, 0, 0 | 3.2 (0) | NA (NA) — No subjects in this treatment group continuing surgery past this time point. | NA (NA) — No subjects in this treatment group continuing surgery past this time point. | NA (NA) — No subjects in this treatment group continuing surgery past this time point.
Statistical Analysis 1: Comparison: Balanced Salt Solution (BSS) vs OMS302 Solution; Test type: Superiority or Other; p = 0.0000, repeated measures model — Repeated measures model includes treatment (OMS302, ketorolac tromethamine, and vehicle), time-point and LOCS II grade as covariates; All data time points collected used in the analysis; least-squares mean difference = 0.9, 95% CI [0.6 to 1.1], Standard Error of Mean 0.1 — OMS302 - Vehicle (BSS)
Statistical Analysis 2: Comparison: OMS302 Anti-inflammatory Solution (KE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.0000, repeated measures model — [p-value comment as in outcome 1, analysis 1]; OMS302 - ketorolac tromethamine; least-squares mean difference = 0.7, 95% CI [0.5 to 0.9], Standard Error of Mean 0.1

2. Primary Outcome: Ocular Pain Visual Analog Scale (VAS) Score (mm) Within 12 Hours Postoperatively
Description: For the primary analysis of this endpoint, only the results on the day of operation at 2, 4, 6, 8 and 10-12 hours were utilized. The VAS scores (where 0 = no pain and 100 = worst possible pain) were summarized by treatment group and time point. Repeated measures analyses of variance were used to test for differences in postoperative ocular pain. The repeated measures model included VAS pain score as the response variable and treatment (OMS302, phenylephrine hydrochloride (PE), and vehicle), time point (as a categorical variable) and the stratification factor LOCS II grade as predictor variables. A generalized estimating equation (GEE) approach with an AR(1) working correlation structure was used.
Time Frame: through 12 hours post-surgery
Population: Subjects with postoperative VAS scores.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Balanced Salt Solution (BSS) | OMS302 Mydriatic Solution (PE) | OMS302 Anti-inflammatory Solution (KE) | OMS302 Solution
Number analyzed (Participants) | 56 | 56 | 55 | 55
units on a scale
  2 hours post-surgery | 8.6 (14.7) | 9.4 (16.8) | 4.1 (12.7) | 5.3 (11.8)
  4 hours post-surgery | 10.9 (19.3) | 10.5 (16.9) | 4.8 (12.3) | 5.9 (12.4)
  6 hours post-surgery | 10.5 (17.2) | 9.5 (14.9) | 4.3 (10.9) | 3.9 (8.6)
  8 hours post-surgery | 8.9 (14.7) | 12.2 (16.9) | 4.0 (11.0) | 4.0 (10.5)
  10-12 hours post-surgery | 10.3 (18.3) | 11.8 (17.1) | 3.4 (9.2) | 4.7 (13.4)
Statistical Analysis 1: Comparison: Balanced Salt Solution (BSS) vs OMS302 Solution; Test type: Superiority or Other; p = 0.0421, repeated measures model — Repeated measures model includes treatment (OMS302, PE and vehicle), time point and LOCS II grade as covariates; least-squares mean difference = -4.6, 95% CI [-8.9 to -0.2], Standard Error of Mean 2.2 — OMS302 - Vehicle (BSS)
Statistical Analysis 2: Comparison: OMS302 Mydriatic Solution (PE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.0093, repeated measures model — Repeated measures model includes treatment (OMS302, PE and vehicle), time point and LOCS II grade as covariates; least-squares mean difference = -5.9, 95% CI [-10.3 to -1.5], Standard Error of Mean 2.2 — OMS302 - PE

3. Secondary Outcome: Ocular Symptoms Using Numerical Rating System - Tearing, Two Hours Post-Surgery
Description: The ocular symptom outcomes were based on Ocular Pain and Symptoms Numerical Ordinal Scale (Numerical Rating System - NRS) at each time point for each assessment (tearing, photophobia, eye discharge, itching, foreign body sensation, and haziness). Treatment comparisons were performed using a Cochran-Mantel- Haenszel (CMH) test adjusting for the stratification factor LOCS II grade.
Time Frame: Two hours
Population: Subjects with scores at time point.
Measure: Number; unit: participants
Arm/Group | Balanced Salt Solution (BSS) | OMS302 Mydriatic Solution (PE) | OMS302 Anti-inflammatory Solution (KE) | OMS302 Solution
Number analyzed (Participants) | 56 | 56 | 55 | 54
participants
  None | 41 | 34 | 48 | 35
  Mild | 12 | 13 | 6 | 14
  Moderate | 3 | 7 | 0 | 4
  Severe | 0 | 2 | 1 | 1
Statistical Analysis 1: Comparison: Balanced Salt Solution (BSS) vs OMS302 Solution; Test type: Superiority or Other; p = 0.630, Cochran-Mantel-Haenszel — Treatment comparisons between OMS302 and each of the other three groups are based on Cochran-Mantel-Haenszel test adjusting for the LOCS II grade group
Statistical Analysis 2: Comparison: OMS302 Mydriatic Solution (PE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.769, Cochran-Mantel-Haenszel — [p-value comment as in outcome 3, analysis 1]
Statistical Analysis 3: Comparison: OMS302 Anti-inflammatory Solution (KE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.025, Cochran-Mantel-Haenszel — [p-value comment as in outcome 3, analysis 1]

4. Secondary Outcome: Ocular Symptoms Using Numerical Rating System - Tearing, Six Hours Post-Surgery
Description: The ocular symptom outcomes were based on Ocular Pain and Symptoms Numerical Ordinal Scale (Numerical Rating System - NRS) at each time point for each assessment (tearing, photophobia, eye discharge, itching, foreign body sensation, and haziness). Treatment comparisons were performed using a Cochran-Mantel-Haenszel (CMH) test adjusting for the stratification factor LOCS II grade.
Time Frame: Six hours
Population: Subjects with scores at time point.
Measure: Number; unit: participants
Arm/Group | Balanced Salt Solution (BSS) | OMS302 Mydriatic Solution (PE) | OMS302 Anti-inflammatory Solution (KE) | OMS302 Solution
Number analyzed (Participants) | 54 | 53 | 50 | 50
participants
  None | 34 | 29 | 43 | 35
  Mild | 12 | 15 | 6 | 13
  Moderate | 7 | 6 | 1 | 1
  Severe | 1 | 3 | 0 | 1
Statistical Analysis 1: Comparison: Balanced Salt Solution (BSS) vs OMS302 Solution; Test type: Superiority or Other; p = 0.229, Cochran-Mantel-Haenszel — [p-value comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: OMS302 Mydriatic Solution (PE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.162, Cochran-Mantel-Haenszel — [p-value comment as in outcome 3, analysis 1]
Statistical Analysis 3: Comparison: OMS302 Anti-inflammatory Solution (KE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.226, Cochran-Mantel-Haenszel — [p-value comment as in outcome 3, analysis 1]

5. Secondary Outcome: Ocular Symptoms Using Numerical Rating System - Tearing, One Day Post-Surgery
Description: as for outcome 4
Time Frame: One day
Population: Subjects with scores at time point.
Measure: Number; unit: participants
Arm/Group | Balanced Salt Solution (BSS) | OMS302 Mydriatic Solution (PE) | OMS302 Anti-inflammatory Solution (KE) | OMS302 Solution
Number analyzed (Participants) | 56 | 55 | 55 | 54
participants
  None | 34 | 29 | 48 | 42
  Mild | 15 | 19 | 6 | 10
  Moderate | 5 | 4 | 1 | 1
  Severe | 2 | 3 | 0 | 1
Statistical Analysis 1: Comparison: Balanced Salt Solution (BSS) vs OMS302 Solution; Test type: Superiority or Other; p = 0.177, Cochran-Mantel-Haenszel — [p-value comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: OMS302 Mydriatic Solution (PE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.051, Cochran-Mantel-Haenszel — [p-value comment as in outcome 3, analysis 1]
Statistical Analysis 3: Comparison: OMS302 Anti-inflammatory Solution (KE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.497, Cochran-Mantel-Haenszel — [p-value comment as in outcome 3, analysis 1]

6. Secondary Outcome: Ocular Symptoms Using Numerical Rating System - Tearing, Two Days Post-Surgery
Description: as for outcome 3
Time Frame: Two days
Population: Subjects with scores at time point.
Measure: Number; unit: participants
Arm/Group | Balanced Salt Solution (BSS) | OMS302 Mydriatic Solution (PE) | OMS302 Anti-inflammatory Solution (KE) | OMS302 Solution
Number analyzed (Participants) | 56 | 55 | 55 | 55
participants
  None | 37 | 30 | 47 | 41
  Mild | 18 | 18 | 7 | 12
  Moderate | 1 | 6 | 0 | 1
  Severe | 0 | 1 | 1 | 1
Statistical Analysis 1: Comparison: Balanced Salt Solution (BSS) vs OMS302 Solution; Test type: Superiority or Other; p = 0.480, Cochran-Mantel-Haenszel — [p-value comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: OMS302 Mydriatic Solution (PE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.090, Cochran-Mantel-Haenszel — [p-value comment as in outcome 3, analysis 1]
Statistical Analysis 3: Comparison: OMS302 Anti-inflammatory Solution (KE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.439, Cochran-Mantel-Haenszel — [p-value comment as in outcome 3, analysis 1]

7. Secondary Outcome: Ocular Symptoms Using Numerical Rating System - Tearing, Seven Days Post-Surgery
Description: as for outcome 3
Time Frame: Seven days
Population: Subjects with scores at time point.
Measure: Number; unit: participants
Arm/Group | Balanced Salt Solution (BSS) | OMS302 Mydriatic Solution (PE) | OMS302 Anti-inflammatory Solution (KE) | OMS302 Solution
Number analyzed (Participants) | 53 | 56 | 53 | 55
participants
  None | 39 | 33 | 46 | 40
  Mild | 13 | 21 | 5 | 13
  Moderate | 1 | 1 | 2 | 1
  Severe | 0 | 1 | 0 | 1
Statistical Analysis 1: Comparison: Balanced Salt Solution (BSS) vs OMS302 Solution; Test type: Superiority or Other; p = 0.812, Cochran-Mantel-Haenszel — [p-value comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: OMS302 Mydriatic Solution (PE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.480, Cochran-Mantel-Haenszel — [p-value comment as in outcome 3, analysis 1]
Statistical Analysis 3: Comparison: OMS302 Anti-inflammatory Solution (KE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.160, Cochran-Mantel-Haenszel — [p-value comment as in outcome 3, analysis 1]

8. Secondary Outcome: Ocular Symptoms Using Numerical Rating System - Tearing, 14 Days Post-Surgery
Description: as for outcome 3
Time Frame: 14 days
Population: Subjects with scores at time point.
Measure: Number; unit: participants
Arm/Group | Balanced Salt Solution (BSS) | OMS302 Mydriatic Solution (PE) | OMS302 Anti-inflammatory Solution (KE) | OMS302 Solution
Number analyzed (Participants) | 55 | 55 | 54 | 53
participants
  None | 44 | 45 | 51 | 42
  Mild | 7 | 10 | 3 | 11
  Moderate | 4 | 0 | 0 | 0
Statistical Analysis 1: Comparison: Balanced Salt Solution (BSS) vs OMS302 Solution; Test type: Superiority or Other; p = 0.085, Cochran-Mantel-Haenszel — [p-value comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: OMS302 Mydriatic Solution (PE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.742, Cochran-Mantel-Haenszel — [p-value comment as in outcome 3, analysis 1]
Statistical Analysis 3: Comparison: OMS302 Anti-inflammatory Solution (KE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.021, Cochran-Mantel-Haenszel — [p-value comment as in outcome 3, analysis 1]

9. Secondary Outcome: Ocular Symptoms Using Numerical Rating System - Tearing, 30 Days Post-Surgery/ Early Termination
Description: as for outcome 3
Time Frame: up to 30 days
Population: Subjects with scores at time point.
Measure: Number; unit: participants
Arm/Group | Balanced Salt Solution (BSS) | OMS302 Mydriatic Solution (PE) | OMS302 Anti-inflammatory Solution (KE) | OMS302 Solution
Number analyzed (Participants) | 55 | 54 | 54 | 53
participants
  None | 43 | 44 | 51 | 49
  Mild | 11 | 9 | 3 | 3
  Moderate | 1 | 1 | 0 | 1
Statistical Analysis 1: Comparison: Balanced Salt Solution (BSS) vs OMS302 Solution; Test type: Superiority or Other; p = 0.081, Cochran-Mantel-Haenszel — [p-value comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: OMS302 Mydriatic Solution (PE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.202, Cochran-Mantel-Haenszel — [p-value comment as in outcome 3, analysis 1]
Statistical Analysis 3: Comparison: OMS302 Anti-inflammatory Solution (KE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.606, Cochran-Mantel-Haenszel — [p-value comment as in outcome 3, analysis 1]

10. Secondary Outcome: Ocular Symptoms Using Numerical Rating System - Photophobia Two Hours Post-Surgery
Description: as for outcome 3
Time Frame: Two hours
Population: Subjects with scores at time point.
Measure: Number; unit: participants
Arm/Group | Balanced Salt Solution (BSS) | OMS302 Mydriatic Solution (PE) | OMS302 Anti-inflammatory Solution (KE) | OMS302 Solution
Number analyzed (Participants) | 56 | 56 | 55 | 54
participants
  None | 37 | 27 | 36 | 32
  Mild | 13 | 22 | 13 | 16
  Moderate | 4 | 3 | 6 | 4
  Severe | 2 | 4 | 0 | 2
Statistical Analysis 1: Comparison: Balanced Salt Solution (BSS) vs OMS302 Solution; Test type: Superiority or Other; p = 0.893, Cochran-Mantel-Haenszel — Treatment comparisons between OMS302 and each of the other three groups are based on Cochran-Mantel- Haenszel test adjusting for the LOCS II grade group
Statistical Analysis 2: Comparison: OMS302 Mydriatic Solution (PE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.553, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]
Statistical Analysis 3: Comparison: OMS302 Anti-inflammatory Solution (KE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.412, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]

11. Secondary Outcome: Ocular Symptoms Using Numerical Rating System - Photophobia Six Hours Post-Surgery
Description: as for outcome 3
Time Frame: Six hours
Population: Subjects with scores at time point.
Measure: Number; unit: participants
Arm/Group | Balanced Salt Solution (BSS) | OMS302 Mydriatic Solution (PE) | OMS302 Anti-inflammatory Solution (KE) | OMS302 Solution
Number analyzed (Participants) | 53 | 53 | 49 | 50
participants
  None | 26 | 29 | 33 | 29
  Mild | 17 | 16 | 12 | 18
  Moderate | 7 | 7 | 4 | 1
  Severe | 3 | 1 | 0 | 2
Statistical Analysis 1: Comparison: Balanced Salt Solution (BSS) vs OMS302 Solution; Test type: Superiority or Other; p = 0.186, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]
Statistical Analysis 2: Comparison: OMS302 Mydriatic Solution (PE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.191, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]
Statistical Analysis 3: Comparison: OMS302 Anti-inflammatory Solution (KE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.167, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]

12. Secondary Outcome: Ocular Symptoms Using Numerical Rating System - Photophobia One Day Post-Surgery
Description: as for outcome 3
Time Frame: One day
Population: Subjects with scores at time point.
Measure: Number; unit: participants
Arm/Group | Balanced Salt Solution (BSS) | OMS302 Mydriatic Solution (PE) | OMS302 Anti-inflammatory Solution (KE) | OMS302 Solution
Number analyzed (Participants) | 56 | 55 | 55 | 54
participants
  None | 20 | 16 | 36 | 23
  Mild | 19 | 22 | 16 | 20
  Moderate | 13 | 11 | 2 | 9
  Severe | 4 | 6 | 1 | 2
Statistical Analysis 1: Comparison: Balanced Salt Solution (BSS) vs OMS302 Solution; Test type: Superiority or Other; p = 0.663, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]
Statistical Analysis 2: Comparison: OMS302 Mydriatic Solution (PE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.326, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]
Statistical Analysis 3: Comparison: OMS302 Anti-inflammatory Solution (KE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.045, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]

13. Secondary Outcome: Ocular Symptoms Using Numerical Rating System - Photophobia Two Days Post-Surgery
Description: as for outcome 3
Time Frame: Two days
Population: Subjects with scores at time point.
Measure: Number; unit: participants
Arm/Group | Balanced Salt Solution (BSS) | OMS302 Mydriatic Solution (PE) | OMS302 Anti-inflammatory Solution (KE) | OMS302 Solution
Number analyzed (Participants) | 56 | 55 | 55 | 55
participants
  None | 26 | 23 | 34 | 19
  Mild | 18 | 24 | 13 | 23
  Moderate | 12 | 4 | 5 | 9
  Severe | 0 | 4 | 3 | 4
Statistical Analysis 1: Comparison: Balanced Salt Solution (BSS) vs OMS302 Solution; Test type: Superiority or Other; p = 0.106, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]
Statistical Analysis 2: Comparison: OMS302 Mydriatic Solution (PE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.519, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]
Statistical Analysis 3: Comparison: OMS302 Anti-inflammatory Solution (KE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.039, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]

14. Secondary Outcome: Ocular Symptoms Using Numerical Rating System - Photophobia Seven Days Post-Surgery
Description: as for outcome 3
Time Frame: Seven days
Population: Subjects with scores at time point.
Measure: Number; unit: participants
Arm/Group | Balanced Salt Solution (BSS) | OMS302 Mydriatic Solution (PE) | OMS302 Anti-inflammatory Solution (KE) | OMS302 Solution
Number analyzed (Participants) | 53 | 56 | 53 | 55
participants
  None | 30 | 31 | 37 | 37
  Mild | 18 | 16 | 11 | 12
  Moderate | 4 | 8 | 3 | 1
  Severe | 1 | 1 | 2 | 5
Statistical Analysis 1: Comparison: Balanced Salt Solution (BSS) vs OMS302 Solution; Test type: Superiority or Other; p = 0.100, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]
Statistical Analysis 2: Comparison: OMS302 Mydriatic Solution (PE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.029, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]
Statistical Analysis 3: Comparison: OMS302 Anti-inflammatory Solution (KE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.525, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]

15. Secondary Outcome: Ocular Symptoms Using Numerical Rating System - Photophobia 14 Days Post-Surgery
Description: as for outcome 3
Time Frame: 14 days
Population: Subjects with scores at time point.
Measure: Number; unit: participants
Arm/Group | Balanced Salt Solution (BSS) | OMS302 Mydriatic Solution (PE) | OMS302 Anti-inflammatory Solution (KE) | OMS302 Solution
Number analyzed (Participants) | 55 | 55 | 54 | 53
participants
  None | 43 | 35 | 42 | 39
  Mild | 10 | 18 | 9 | 12
  Moderate | 2 | 2 | 3 | 1
  Severe | 0 | 0 | 0 | 1
Statistical Analysis 1: Comparison: Balanced Salt Solution (BSS) vs OMS302 Solution; Test type: Superiority or Other; p = 0.642, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]
Statistical Analysis 2: Comparison: OMS302 Mydriatic Solution (PE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.442, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]
Statistical Analysis 3: Comparison: OMS302 Anti-inflammatory Solution (KE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.467, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]

16. Secondary Outcome: Ocular Symptoms Using Numerical Rating System - Photophobia 30 Days Post-Surgery /Early Termination
Description: as for outcome 3
Time Frame: Up to 30 days
Population: Subjects with scores at time point.
Measure: Number; unit: participants
Arm/Group | Balanced Salt Solution (BSS) | OMS302 Mydriatic Solution (PE) | OMS302 Anti-inflammatory Solution (KE) | OMS302 Solution
Number analyzed (Participants) | 55 | 54 | 54 | 53
participants
  None | 44 | 36 | 42 | 40
  Mild | 10 | 17 | 12 | 10
  Moderate | 1 | 1 | 0 | 2
  Severe | 0 | 0 | 0 | 1
Statistical Analysis 1: Comparison: Balanced Salt Solution (BSS) vs OMS302 Solution; Test type: Superiority or Other; p = 0.695, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]
Statistical Analysis 2: Comparison: OMS302 Mydriatic Solution (PE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.355, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]
Statistical Analysis 3: Comparison: OMS302 Anti-inflammatory Solution (KE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.369, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]

17. Secondary Outcome: Ocular Symptoms Using Numerical Rating System - Eye Discharge 2 Hours Post-Surgery
Description: as for outcome 3
Time Frame: Two hours
Population: Subjects with scores at time point.
Measure: Number; unit: participants
Groups:
- Solution: Balanced Salt Solution (BSS)
  Balanced Salt Solution (BSS)
Arm/Group | Solution | OMS302 Mydriatic Solution (PE) | OMS302 Anti-inflammatory Solution (KE) | OMS302 Solution
Number analyzed (Participants) | 56 | 56 | 55 | 54
participants
  None | 55 | 50 | 52 | 48
  Mild | 1 | 6 | 2 | 4
  Moderate | 0 | 0 | 0 | 2
  Severe | 0 | 0 | 1 | 0
Statistical Analysis 1: Comparison: Solution vs OMS302 Solution; Test type: Superiority or Other; p = 0.124, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]
Statistical Analysis 2: Comparison: OMS302 Mydriatic Solution (PE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.298, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]
Statistical Analysis 3: Comparison: OMS302 Anti-inflammatory Solution (KE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.291, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]

18. Secondary Outcome: Ocular Symptoms Using Numerical Rating System - Eye Discharge Six Hours Post-Surgery
Description: as for outcome 3
Time Frame: Six hours
Population: Subjects with scores at time point.
Measure: Number; unit: participants
Arm/Group | Balanced Salt Solution (BSS) | OMS302 Mydriatic Solution (PE) | OMS302 Anti-inflammatory Solution (KE) | OMS302 Solution
Number analyzed (Participants) | 54 | 53 | 50 | 50
participants
  None | 44 | 49 | 41 | 43
  Mild | 7 | 1 | 8 | 5
  Moderate | 3 | 3 | 1 | 2
  Severe | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: Balanced Salt Solution (BSS) vs OMS302 Solution; Test type: Superiority or Other; p = 0.825, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]
Statistical Analysis 2: Comparison: OMS302 Mydriatic Solution (PE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.211, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]
Statistical Analysis 3: Comparison: OMS302 Anti-inflammatory Solution (KE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.589, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]

19. Secondary Outcome: Ocular Symptoms Using Numerical Rating System - Eye Discharge One Day Post-Surgery
Description: as for outcome 3
Time Frame: One day
Population: Subjects with scores at time point.
Measure: Number; unit: participants
Arm/Group | Balanced Salt Solution (BSS) | OMS302 Mydriatic Solution (PE) | OMS302 Anti-inflammatory Solution (KE) | OMS302 Solution
Number analyzed (Participants) | 56 | 55 | 55 | 54
participants
  None | 48 | 45 | 48 | 50
  Mild | 7 | 9 | 6 | 4
  Moderate | 0 | 1 | 1 | 0
  Severe | 1 | 0 | 0 | 0
Statistical Analysis 1: Comparison: Balanced Salt Solution (BSS) vs OMS302 Solution; Test type: Superiority or Other; p = 0.401, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]
Statistical Analysis 2: Comparison: OMS302 Mydriatic Solution (PE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.200, Chi-squared, Corrected — [p-value comment as in outcome 10, analysis 1]
Statistical Analysis 3: Comparison: OMS302 Anti-inflammatory Solution (KE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.478, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]

20. Secondary Outcome: Ocular Symptoms Using Numerical Rating System - Eye Discharge Two Days Post-Surgery
Description: as for outcome 3
Time Frame: Two days
Population: Subjects with scores at time point.
Measure: Number; unit: participants
Arm/Group | Balanced Salt Solution (BSS) | OMS302 Mydriatic Solution (PE) | OMS302 Anti-inflammatory Solution (KE) | OMS302 Solution
Number analyzed (Participants) | 56 | 55 | 55 | 55
participants
  None | 52 | 48 | 46 | 49
  Mild | 3 | 7 | 8 | 5
  Moderate | 1 | 0 | 0 | 1
  Severe | 0 | 0 | 1 | 0
Statistical Analysis 1: Comparison: Balanced Salt Solution (BSS) vs OMS302 Solution; Test type: Superiority or Other; p = 0.758, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]
Statistical Analysis 2: Comparison: OMS302 Mydriatic Solution (PE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.521, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]
Statistical Analysis 3: Comparison: OMS302 Anti-inflammatory Solution (KE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.432, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]

21. Secondary Outcome: Ocular Symptoms Using Numerical Rating System - Eye Discharge Seven Days Post-Surgery
Description: as for outcome 3
Time Frame: Seven days
Population: Subjects with scores at time point.
Measure: Number; unit: participants
Arm/Group | Balanced Salt Solution (BSS) | OMS302 Mydriatic Solution (PE) | OMS302 Anti-inflammatory Solution (KE) | OMS302 Solution
Number analyzed (Participants) | 53 | 56 | 53 | 55
participants
  None | 49 | 52 | 52 | 52
  Mild | 4 | 4 | 1 | 1
  Moderate | 0 | 0 | 0 | 2
  Severe | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: Balanced Salt Solution (BSS) vs OMS302 Solution; Test type: Superiority or Other; p = 0.148, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]
Statistical Analysis 2: Comparison: OMS302 Mydriatic Solution (PE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.156, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]
Statistical Analysis 3: Comparison: OMS302 Anti-inflammatory Solution (KE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.381, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]

22. Secondary Outcome: Ocular Symptoms Using Numerical Rating System - Eye Discharge 14 Days Post-Surgery
Description: as for outcome 3
Time Frame: 14 days
Population: Subjects with scores at time point.
Measure: Number; unit: participants
Arm/Group | Balanced Salt Solution (BSS) | OMS302 Mydriatic Solution (PE) | OMS302 Anti-inflammatory Solution (KE) | OMS302 Solution
Number analyzed (Participants) | 55 | 55 | 54 | 53
participants
  None | 52 | 51 | 53 | 49
  Mild | 3 | 4 | 1 | 4
  Moderate | 0 | 0 | 0 | 0
  Severe | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: Balanced Salt Solution (BSS) vs OMS302 Solution; Test type: Superiority or Other; p = 0.646, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]
Statistical Analysis 2: Comparison: OMS302 Mydriatic Solution (PE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.950, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]
Statistical Analysis 3: Comparison: OMS302 Anti-inflammatory Solution (KE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.160, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]

23. Secondary Outcome: Ocular Symptoms Using Numerical Rating System - Eye Discharge 30 Days Post-Surgery/Early Termination
Description: as for outcome 3
Time Frame: Up to 30 days
Population: Subjects with scores at time point.
Measure: Number; unit: participants
Arm/Group | Balanced Salt Solution (BSS) | OMS302 Mydriatic Solution (PE) | OMS302 Anti-inflammatory Solution (KE) | OMS302 Solution
Number analyzed (Participants) | 55 | 54 | 54 | 53
participants
  None | 52 | 52 | 53 | 50
  Mild | 3 | 2 | 1 | 3
  Moderate | 0 | 0 | 0 | 0
  Severe | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: Balanced Salt Solution (BSS) vs OMS302 Solution; Test type: Superiority or Other; p = 1.000, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]
Statistical Analysis 2: Comparison: OMS302 Mydriatic Solution (PE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.667, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]
Statistical Analysis 3: Comparison: OMS302 Anti-inflammatory Solution (KE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.303, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]

24. Secondary Outcome: Ocular Symptoms Using Numerical Rating System - Itching Two Hours Post-Surgery
Description: as for outcome 3
Time Frame: Two hours
Population: Subjects with scores at time point.
Measure: Number; unit: participants
Arm/Group | Balanced Salt Solution (BSS) | OMS302 Mydriatic Solution (PE) | OMS302 Anti-inflammatory Solution (KE) | OMS302 Solution
Number analyzed (Participants) | 56 | 56 | 55 | 54
participants
  None | 49 | 48 | 45 | 47
  Mild | 5 | 7 | 9 | 6
  Moderate | 1 | 1 | 1 | 1
  Severe | 1 | 0 | 0 | 0
Statistical Analysis 1: Comparison: Balanced Salt Solution (BSS) vs OMS302 Solution; Test type: Superiority or Other; p = 0.789, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]
Statistical Analysis 2: Comparison: OMS302 Mydriatic Solution (PE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.977, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]
Statistical Analysis 3: Comparison: OMS302 Anti-inflammatory Solution (KE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.336, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]

25. Secondary Outcome: Ocular Symptoms Using Numerical Rating System - Itching 6 Hours Post-Surgery
Description: as for outcome 3
Time Frame: Six hours
Population: Subjects with scores at time point.
Measure: Number; unit: participants
Arm/Group | Balanced Salt Solution (BSS) | OMS302 Mydriatic Solution (PE) | OMS302 Anti-inflammatory Solution (KE) | OMS302 Solution
Number analyzed (Participants) | 54 | 53 | 49 | 50
participants
  None | 44 | 43 | 39 | 43
  Mild | 7 | 9 | 10 | 6
  Moderate | 3 | 1 | 0 | 1
  Severe | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: Balanced Salt Solution (BSS) vs OMS302 Solution; Test type: Superiority or Other; p = 0.632, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]
Statistical Analysis 2: Comparison: OMS302 Mydriatic Solution (PE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.778, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]
Statistical Analysis 3: Comparison: OMS302 Anti-inflammatory Solution (KE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.336, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]

26. Secondary Outcome: Ocular Symptoms Using Numerical Rating System - Itching One Day Post-Surgery
Description: as for outcome 3
Time Frame: One day
Population: Subjects with scores at time point.
Measure: Number; unit: participants
Arm/Group | Balanced Salt Solution (BSS) | OMS302 Mydriatic Solution (PE) | OMS302 Anti-inflammatory Solution (KE) | OMS302 Solution
Number analyzed (Participants) | 56 | 55 | 55 | 54
participants
  None | 45 | 49 | 49 | 46
  Mild | 10 | 6 | 6 | 6
  Moderate | 1 | 0 | 0 | 2
  Severe | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: Balanced Salt Solution (BSS) vs OMS302 Solution; Test type: Superiority or Other; p = 0.528, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]
Statistical Analysis 2: Comparison: OMS302 Mydriatic Solution (PE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.362, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]
Statistical Analysis 3: Comparison: OMS302 Anti-inflammatory Solution (KE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.353, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]

27. Secondary Outcome: Ocular Symptoms Using Numerical Rating System - Itching Two Days Post-Surgery
Description: as for outcome 3
Time Frame: Two days
Population: Subjects with scores at time point.
Measure: Number; unit: participants
Arm/Group | Balanced Salt Solution (BSS) | OMS302 Mydriatic Solution (PE) | OMS302 Anti-inflammatory Solution (KE) | OMS302 Solution
Number analyzed (Participants) | 56 | 55 | 55 | 55
participants
  None | 45 | 44 | 46 | 41
  Mild | 11 | 10 | 9 | 14
  Moderate | 0 | 1 | 0 | 0
  Severe | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: Balanced Salt Solution (BSS) vs OMS302 Solution; Test type: Superiority or Other; p = 0.463, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]
Statistical Analysis 2: Comparison: OMS302 Mydriatic Solution (PE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.406, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]
Statistical Analysis 3: Comparison: OMS302 Anti-inflammatory Solution (KE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.245, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]

28. Secondary Outcome: Ocular Symptoms Using Numerical Rating System - Itching Seven Days Post-Surgery
Description: as for outcome 3
Time Frame: Seven days
Population: Subjects with scores at time point.
Measure: Number; unit: participants
Arm/Group | Balanced Salt Solution (BSS) | OMS302 Mydriatic Solution (PE) | OMS302 Anti-inflammatory Solution (KE) | OMS302 Solution
Number analyzed (Participants) | 53 | 56 | 53 | 55
participants
  None | 39 | 47 | 40 | 42
  Mild | 13 | 9 | 13 | 12
  Moderate | 1 | 0 | 0 | 1
  Severe | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: Balanced Salt Solution (BSS) vs OMS302 Solution; Test type: Superiority or Other; p = 0.945, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]
Statistical Analysis 2: Comparison: OMS302 Mydriatic Solution (PE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.438, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]
Statistical Analysis 3: Comparison: OMS302 Anti-inflammatory Solution (KE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.596, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]

29. Secondary Outcome: Ocular Symptoms Using Numerical Rating System - Itching 14 Days Post-Surgery
Description: as for outcome 3
Time Frame: 14 days
Population: Subjects with scores at time point.
Measure: Number; unit: participants
Arm/Group | Balanced Salt Solution (BSS) | OMS302 Mydriatic Solution (PE) | OMS302 Anti-inflammatory Solution (KE) | OMS302 Solution
Number analyzed (Participants) | 55 | 55 | 54 | 53
participants
  None | 48 | 45 | 44 | 44
  Mild | 6 | 10 | 10 | 8
  Moderate | 1 | 0 | 0 | 1
  Severe | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: Balanced Salt Solution (BSS) vs OMS302 Solution; Test type: Superiority or Other; p = 0.811, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]
Statistical Analysis 2: Comparison: OMS302 Mydriatic Solution (PE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.552, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]
Statistical Analysis 3: Comparison: OMS302 Anti-inflammatory Solution (KE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.549, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]

30. Secondary Outcome: Ocular Symptoms Using Numerical Rating System - Itching 30 Days Post-Surgery/Early Termination
Description: as for outcome 3
Time Frame: Up to 30 days
Population: Subjects with scores at time point.
Measure: Number; unit: participants
Arm/Group | Balanced Salt Solution (BSS) | OMS302 Mydriatic Solution (PE) | OMS302 Anti-inflammatory Solution (KE) | OMS302 Solution
Number analyzed (Participants) | 55 | 54 | 54 | 53
participants
  None | 43 | 46 | 47 | 48
  Mild | 11 | 8 | 7 | 5
  Moderate | 1 | 0 | 0 | 0
  Severe | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: Balanced Salt Solution (BSS) vs OMS302 Solution; Test type: Superiority or Other; p = 0.173, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]
Statistical Analysis 2: Comparison: OMS302 Mydriatic Solution (PE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.362, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]
Statistical Analysis 3: Comparison: OMS302 Anti-inflammatory Solution (KE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.559, Cochran-Mantel-Haenszel

31. Secondary Outcome: Ocular Symptoms Using Numerical Rating System - Foreign Body Sensation Two Hours Post-Surgery
Description: as for outcome 3
Time Frame: Two hours
Population: Subjects with scores at time point.
Measure: Number; unit: participants
Arm/Group | Balanced Salt Solution (BSS) | OMS302 Mydriatic Solution (PE) | OMS302 Anti-inflammatory Solution (KE) | OMS302 Solution
Number analyzed (Participants) | 56 | 56 | 55 | 54
participants
  None | 32 | 26 | 31 | 25
  Mild | 17 | 24 | 20 | 19
  Moderate | 6 | 4 | 3 | 9
  Severe | 1 | 2 | 1 | 1
Statistical Analysis 1: Comparison: Balanced Salt Solution (BSS) vs OMS302 Solution; Test type: Superiority or Other; p = 0.681, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]
Statistical Analysis 2: Comparison: OMS302 Mydriatic Solution (PE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.429, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]
Statistical Analysis 3: Comparison: OMS302 Anti-inflammatory Solution (KE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.306, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]

32. Secondary Outcome: Ocular Symptoms Using Numerical Rating System - Foreign Body Sensation Six Hours Post-Surgery
Description: as for outcome 3
Time Frame: Six hours
Population: Subjects with scores at time point.
Measure: Number; unit: participants
Arm/Group | Balanced Salt Solution (BSS) Solution | OMS302 Mydriatic Solution (PE) | OMS302 Anti-inflammatory Solution (KE) | OMS302 Solution
Number analyzed (Participants) | 54 | 53 | 49 | 50
participants
  None | 26 | 31 | 31 | 34
  Mild | 19 | 16 | 16 | 10
  Moderate | 8 | 4 | 2 | 5
  Severe | 1 | 2 | 0 | 1
Statistical Analysis 1: Comparison: Balanced Salt Solution (BSS) Solution vs OMS302 Solution; Test type: Superiority or Other; p = 0.226, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]
Statistical Analysis 2: Comparison: OMS302 Mydriatic Solution (PE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.602, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]
Statistical Analysis 3: Comparison: OMS302 Anti-inflammatory Solution (KE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.290, Cochran-Mantel-Haenszel

33. Secondary Outcome: Ocular Symptoms Using Numerical Rating System - Foreign Body Sensation One Day Post-Surgery
Description: as for outcome 3
Time Frame: One day
Population: Subjects with scores at time point.
Measure: Number; unit: participants
Arm/Group | Balanced Salt Solution (BSS) Solution | OMS302 Mydriatic Solution (PE) | OMS302 Anti-inflammatory Solution (KE) | OMS302 Solution
Number analyzed (Participants) | 56 | 55 | 55 | 54
participants
  None | 36 | 25 | 37 | 35
  Mild | 13 | 25 | 16 | 16
  Moderate | 7 | 5 | 2 | 2
  Severe | 0 | 0 | 0 | 1
Statistical Analysis 1: Comparison: Balanced Salt Solution (BSS) Solution vs OMS302 Solution; Test type: Superiority or Other; p = 0.244, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]
Statistical Analysis 2: Comparison: OMS302 Mydriatic Solution (PE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.122, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]
Statistical Analysis 3: Comparison: OMS302 Anti-inflammatory Solution (KE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.790, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]

34. Secondary Outcome: Ocular Symptoms Using Numerical Rating System - Foreign Body Sensation Two Days Post-Surgery
Description: as for outcome 3
Time Frame: Two days
Population: Subjects with scores at time point.
Measure: Number; unit: participants
Arm/Group | Balanced Salt Solution (BSS) | OMS302 Mydriatic Solution (PE) | OMS302 Anti-inflammatory Solution (KE) | OMS302 Solution
Number analyzed (Participants) | 56 | 55 | 55 | 55
participants
  None | 37 | 39 | 38 | 35
  Mild | 16 | 11 | 15 | 15
  Moderate | 3 | 3 | 1 | 5
  Severe | 0 | 2 | 1 | 0
Statistical Analysis 1: Comparison: Balanced Salt Solution (BSS) vs OMS302 Solution; Test type: Superiority or Other; p = 0.752, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]
Statistical Analysis 2: Comparison: OMS302 Mydriatic Solution (PE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.355, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]
Statistical Analysis 3: Comparison: OMS302 Anti-inflammatory Solution (KE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.292, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]

35. Secondary Outcome: Ocular Symptoms Using Numerical Rating System - Foreign Body Sensation Seven Days Post-Surgery 7 Days
Description: as for outcome 3
Time Frame: Seven days
Population: Subjects with scores at time point.
Measure: Number; unit: participants
Arm/Group | Balanced Salt Solution (BSS) | OMS302 Mydriatic Solution (PE) | OMS302 Anti-inflammatory Solution (KE) | OMS302 Solution
Number analyzed (Participants) | 53 | 56 | 53 | 55
participants
  None | 27 | 32 | 34 | 37
  Mild | 23 | 17 | 17 | 15
  Moderate | 3 | 5 | 2 | 2
  Severe | 0 | 2 | 0 | 1
Statistical Analysis 1: Comparison: Balanced Salt Solution (BSS) vs OMS302 Solution; Test type: Superiority or Other; p = 0.228, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]
Statistical Analysis 2: Comparison: OMS302 Mydriatic Solution (PE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.564, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]
Statistical Analysis 3: Comparison: OMS302 Anti-inflammatory Solution (KE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.755, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]

36. Secondary Outcome: Ocular Symptoms Using Numerical Rating System - Foreign Body Sensation 14 Days Post-Surgery
Description: as for outcome 3
Time Frame: 14 days
Population: Subjects with scores at time point.
Measure: Number; unit: participants
Arm/Group | Balanced Salt Solution (BSS) | OMS302 Mydriatic Solution (PE) | OMS302 Anti-inflammatory Solution (KE) | OMS302 Solution
Number analyzed (Participants) | 55 | 55 | 54 | 53
participants
  None | 31 | 38 | 36 | 42
  Mild | 23 | 16 | 16 | 9
  Moderate | 1 | 1 | 1 | 2
  Severe | 0 | 0 | 1 | 0
Statistical Analysis 1: Comparison: Balanced Salt Solution (BSS) vs OMS302 Solution; Test type: Superiority or Other; p = 0.018, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]
Statistical Analysis 2: Comparison: OMS302 Mydriatic Solution (PE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.292, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]
Statistical Analysis 3: Comparison: OMS302 Anti-inflammatory Solution (KE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.298, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]

37. Secondary Outcome: Ocular Symptoms Using Numerical Rating System - Foreign Body Sensation 30 Days Post-Surgery/Early Termination
Description: as for outcome 3
Time Frame: Up to 30 days
Population: Subjects with scores at time point.
Measure: Number; unit: participants
Arm/Group | Balanced Salt Solution (BSS) | OMS302 Mydriatic Solution (PE) | OMS302 Anti-inflammatory Solution (KE) | OMS302 Solution
Number analyzed (Participants) | 55 | 54 | 54 | 53
participants
  None | 41 | 44 | 40 | 46
  Mild | 12 | 10 | 14 | 6
  Moderate | 2 | 0 | 0 | 1
  Severe | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: Balanced Salt Solution (BSS) vs OMS302 Solution; Test type: Superiority or Other; p = 0.271, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]
Statistical Analysis 2: Comparison: OMS302 Mydriatic Solution (PE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.345, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]
Statistical Analysis 3: Comparison: OMS302 Anti-inflammatory Solution (KE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.096, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]

38. Secondary Outcome: Ocular Symptoms Using Numerical Rating System - Haziness Two Hours Post-Surgery
Description: as for outcome 3
Time Frame: Two hours
Population: Subjects with scores at time point.
Measure: Number; unit: participants
Arm/Group | Balanced Salt Solution (BSS) | OMS302 Mydriatic Solution (PE) | OMS302 Anti-inflammatory Solution (KE) | OMS302 Solution
Number analyzed (Participants) | 56 | 56 | 55 | 54
participants
  None | 27 | 24 | 28 | 17
  Mild | 21 | 17 | 18 | 25
  Moderate | 6 | 12 | 8 | 10
  Severe | 2 | 3 | 1 | 2
Statistical Analysis 1: Comparison: Balanced Salt Solution (BSS) vs OMS302 Solution; Test type: Superiority or Other; p = 0.320, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]
Statistical Analysis 2: Comparison: OMS302 Mydriatic Solution (PE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.390, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]
Statistical Analysis 3: Comparison: OMS302 Anti-inflammatory Solution (KE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.230, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]

39. Secondary Outcome: Ocular Symptoms Using Numerical Rating System - Haziness Six Hours Post-Surgery
Description: as for outcome 3
Time Frame: Six hours
Population: Subjects with scores at time point.
Measure: Number; unit: participants
Arm/Group | Balanced Salt Solution (BSS) | OMS302 Mydriatic Solution (PE) | OMS302 Anti-inflammatory Solution (KE) | OMS302 Solution
Number analyzed (Participants) | 53 | 53 | 49 | 50
participants
  None | 24 | 20 | 26 | 23
  Mild | 21 | 20 | 13 | 19
  Moderate | 7 | 10 | 10 | 8
  Severe | 1 | 3 | 0 | 0
Statistical Analysis 1: Comparison: Balanced Salt Solution (BSS) vs OMS302 Solution; Test type: Superiority or Other; p = 0.778, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]
Statistical Analysis 2: Comparison: OMS302 Mydriatic Solution (PE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.348, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]
Statistical Analysis 3: Comparison: OMS302 Anti-inflammatory Solution (KE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.477, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]

40. Secondary Outcome: Ocular Symptoms Using Numerical Rating System - Haziness One Day Post-Surgery
Description: as for outcome 3
Time Frame: One day
Population: Subjects with scores at time point.
Measure: Number; unit: participants
Arm/Group | Balanced Salt Solution (BSS) | OMS302 Mydriatic Solution (PE) | OMS302 Anti-inflammatory Solution (KE) | OMS302 Solution
Number analyzed (Participants) | 56 | 55 | 55 | 54
participants
  None | 34 | 29 | 36 | 38
  Mild | 15 | 19 | 17 | 12
  Moderate | 7 | 4 | 2 | 3
  Severe | 0 | 3 | 0 | 1
Statistical Analysis 1: Comparison: Balanced Salt Solution (BSS) vs OMS302 Solution; Test type: Superiority or Other; p = 0.374, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]
Statistical Analysis 2: Comparison: OMS302 Mydriatic Solution (PE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.265, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]
Statistical Analysis 3: Comparison: OMS302 Anti-inflammatory Solution (KE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.555, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]

41. Secondary Outcome: Ocular Symptoms Using Numerical Rating System - Haziness Two Days Post-Surgery
Description: as for outcome 3
Time Frame: Two days
Population: Subjects with scores at time point.
Measure: Number; unit: participants
Arm/Group | Balanced Salt Solution (BSS) | OMS302 Mydriatic Solution (PE) | OMS302 Anti-inflammatory Solution (KE) | OMS302 Solution
Number analyzed (Participants) | 56 | 55 | 55 | 55
participants
  None | 36 | 31 | 39 | 43
  Mild | 19 | 17 | 13 | 8
  Moderate | 1 | 5 | 3 | 4
  Severe | 0 | 2 | 0 | 0
Statistical Analysis 1: Comparison: Balanced Salt Solution (BSS) vs OMS302 Solution; Test type: Superiority or Other; p = 0.031, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]
Statistical Analysis 2: Comparison: OMS302 Mydriatic Solution (PE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.059, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]
Statistical Analysis 3: Comparison: OMS302 Anti-inflammatory Solution (KE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.472, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]

42. Secondary Outcome: Ocular Symptoms Using Numerical Rating System - Haziness Seven Days Post-Surgery
Description: as for outcome 3
Time Frame: Seven days
Population: Subjects with scores at time point.
Measure: Number; unit: participants
Arm/Group | Balanced Salt Solution (BSS) | OMS302 Mydriatic Solution (PE) | OMS302 Anti-inflammatory Solution (KE) | OMS302 Solution
Number analyzed (Participants) | 53 | 56 | 53 | 55
participants
  None | 36 | 33 | 34 | 41
  Mild | 16 | 17 | 18 | 11
  Moderate | 1 | 6 | 1 | 2
  Severe | 0 | 0 | 0 | 1
Statistical Analysis 1: Comparison: Balanced Salt Solution (BSS) vs OMS302 Solution; Test type: Superiority or Other; p = 0.476, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]
Statistical Analysis 2: Comparison: OMS302 Mydriatic Solution (PE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.169, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]
Statistical Analysis 3: Comparison: OMS302 Anti-inflammatory Solution (KE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.310, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]

43. Secondary Outcome: Ocular Symptoms Using Numerical Rating System - Haziness 14 Days Post-Surgery
Description: as for outcome 3
Time Frame: 14 days
Population: Subjects with scores at time point.
Measure: Number; unit: participants
Arm/Group | Balanced Salt Solution (BSS) | OMS302 Mydriatic Solution (PE) | OMS302 Anti-inflammatory Solution (KE) | OMS302 Solution
Number analyzed (Participants) | 55 | 55 | 54 | 53
participants
  None | 39 | 34 | 39 | 47
  Mild | 10 | 16 | 13 | 4
  Moderate | 6 | 5 | 1 | 2
  Severe | 0 | 0 | 1 | 0
Statistical Analysis 1: Comparison: Balanced Salt Solution (BSS) vs OMS302 Solution; Test type: Superiority or Other; p = 0.075, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]
Statistical Analysis 2: Comparison: OMS302 Mydriatic Solution (PE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.005, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]
Statistical Analysis 3: Comparison: OMS302 Anti-inflammatory Solution (KE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.078, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]

44. Secondary Outcome: Ocular Symptoms Using Numerical Rating System - Haziness 30 Days Post-Surgery/Early Termination
Description: as for outcome 3
Time Frame: Up to 30 days
Population: Subjects with scores at time point.
Measure: Number; unit: participants
Arm/Group | Balanced Salt Solution (BSS) | OMS302 Mydriatic Solution (PE) | OMS302 Anti-inflammatory Solution (KE) | OMS302 Solution
Number analyzed (Participants) | 55 | 54 | 54 | 53
participants
  None | 38 | 42 | 44 | 44
  Mild | 14 | 6 | 10 | 7
  Moderate | 3 | 6 | 0 | 2
  Severe | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: Balanced Salt Solution (BSS) vs OMS302 Solution; Test type: Superiority or Other; p = 0.226, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]
Statistical Analysis 2: Comparison: OMS302 Mydriatic Solution (PE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.357, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]
Statistical Analysis 3: Comparison: OMS302 Anti-inflammatory Solution (KE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.291, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]

45. Secondary Outcome: Best Corrected Visual Acuity (BVCA) - Log Score, Baseline
Description: Best-Corrected Visual Acuity (BCVA) was summarized by the Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity log score. For subjects without a score due to inability to read the ETDRS chart, the log score was imputed as 1.6 for the purpose of treatment comparisons. Subjects without a score because the manifest refraction was not completed were excluded from the analysis. Treatment comparisons for BCVA were performed by pairwise Wilcoxon tests.
Time Frame: Baseline
Population: Subjects with scores at time point.
Measure: Mean (Standard Deviation); unit: Log score
Arm/Group | Balanced Salt Solution (BSS) | OMS302 Mydriatic Solution (PE) | OMS302 Anti-inflammatory Solution (KE) | OMS302 Solution
Number analyzed (Participants) | 54 | 55 | 53 | 56
Log score | 0.4 (0.3) | 0.4 (0.2) | 0.4 (0.2) | 0.4 (0.3)
Statistical Analysis 1: Comparison: Balanced Salt Solution (BSS) vs OMS302 Solution; Test type: Superiority or Other; p = 0.172, Wilcoxon rank-sum test — Treatment comparisons between OMS302 and each of the other three groups are based on Wilcoxon rank-sum test
Statistical Analysis 2: Comparison: OMS302 Mydriatic Solution (PE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.547, Wilcoxon rank-sum test — Treatment comparisons between OMS302 and each of the other three groups are based on Wilcoxon rank-sum test
Statistical Analysis 3: Comparison: OMS302 Anti-inflammatory Solution (KE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.921, Wicoxon rank-sum test — Treatment comparisons between OMS302 and each of the other three groups are based on Wilcoxon rank-sum test

46. Secondary Outcome: Best Corrected Visual Acuity (BVCA) - Log Score, Day 1
Description: Best-Corrected Visual Acuity (BCVA) was summarized by the ETDRS visual acuity log score. For subjects without a score due to inability to read the ETDRS chart, the log score was imputed as 1.6 for the purpose of treatment comparisons. Subjects without a score because the manifest refraction was not completed were excluded from the analysis. Treatment comparisons for BCVA were performed by pairwise Wilcoxon tests.
Time Frame: One day
Population: Subjects with scores at time point.
Measure: Mean (Standard Deviation); unit: Log score
Arm/Group | Balanced Salt Solution (BSS) | OMS302 Mydriatic Solution (PE) | OMS302 Anti-inflammatory Solution (KE) | OMS302 Solution
Number analyzed (Participants) | 56 | 55 | 55 | 54
Log score | 0.1 (0.2) | 0.2 (0.3) | 0.2 (0.2) | 0.1 (0.2)
Statistical Analysis 1: Comparison: Balanced Salt Solution (BSS) vs OMS302 Solution; Test type: Superiority or Other; p = 0.701, Wilcoxon rank-sum test — Treatment comparisons between OMS302 and each of the other three groups are based on Wilcoxon rank-sum test
Statistical Analysis 2: Comparison: OMS302 Mydriatic Solution (PE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.089, Wilcoxon rank-sum test — Treatment comparisons between OMS302 and each of the other three groups are based on Wilcoxon rank-sum test
Statistical Analysis 3: Comparison: OMS302 Anti-inflammatory Solution (KE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.095, Wilcoxon rank-sum test — Treatment comparisons between OMS302 and each of the other three groups are based on Wilcoxon rank-sum test

47. Secondary Outcome: Best Corrected Visual Acuity (BVCA) - Log Score, Day 2
Description: as for outcome 46
Time Frame: Two days
Population: Subjects with scores at time point.
Measure: Mean (Standard Deviation); unit: Log score
Arm/Group | Balanced Salt Solution (BSS) | OMS302 Mydriatic Solution (PE) | OMS302 Anti-inflammatory Solution (KE) | OMS302 Solution
Number analyzed (Participants) | 56 | 56 | 55 | 55
Log score | 0.1 (0.2) | 0.2 (0.3) | 0.1 (0.2) | 0.1 (0.1)
Statistical Analysis 1: Comparison: Balanced Salt Solution (BSS) vs OMS302 Solution; Test type: Superiority or Other; p = 0.086, Wilcoxon rank-sum test — Treatment comparisons between OMS302 and each of the other three groups are based on Wilcoxon rank-sum test
Statistical Analysis 2: Comparison: OMS302 Mydriatic Solution (PE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.092, Wicoxon rank-sum test — Treatment comparisons between OMS302 and each of the other three groups are based on Wilcoxon rank-sum test
Statistical Analysis 3: Comparison: OMS302 Anti-inflammatory Solution (KE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.120, Wilcoxon rank-sum test — Treatment comparisons between OMS302 and each of the other three groups are based on Wilcoxon rank-sum test

48. Secondary Outcome: Best Corrected Visual Acuity (BVCA) - Log Score, Day 7
Description: as for outcome 46
Time Frame: Seven days
Population: Subjects with scores at time point.
Measure: Mean (Standard Deviation); unit: Log score
Arm/Group | Balanced Salt Solution (BSS) | OMS302 Mydriatic Solution (PE) | OMS302 Anti-inflammatory Solution (KE) | OMS302 Solution
Number analyzed (Participants) | 56 | 56 | 53 | 55
Log score | 0.1 (0.2) | 0.1 (0.2) | 0.1 (0.1) | 0.1 (0.2)
Statistical Analysis 1: Comparison: Balanced Salt Solution (BSS) vs OMS302 Solution; Test type: Superiority or Other; p = 0.626, Wilcoxon rank-sum test — Treatment comparisons between OMS302 and each of the other three groups are based on Wilcoxon rank-sum test
Statistical Analysis 2: Comparison: OMS302 Mydriatic Solution (PE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.736, Wilcoxon rank-sum test — Treatment comparisons between OMS302 and each of the other three groups are based on Wilcoxon rank-sum test
Statistical Analysis 3: Comparison: OMS302 Anti-inflammatory Solution (KE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.725, Wilcoxon rank-sum test — Treatment comparisons between OMS302 and each of the other three groups are based on Wilcoxon rank-sum test

49. Secondary Outcome: Best Corrected Visual Acuity (BVCA) - Log Score, Day 14
Description: as for outcome 46
Time Frame: 14 days
Population: Subjects with scores at time point.
Measure: Mean (Standard Deviation); unit: Log score
Arm/Group | Balanced Salt Solution (BSS) | OMS302 Mydriatic Solution (PE) | OMS302 Anti-inflammatory Solution (KE) | OMS302 Solution
Number analyzed (Participants) | 55 | 56 | 55 | 53
Log score | 0.1 (0.2) | 0.1 (0.2) | 0.1 (0.2) | 0.1 (0.1)
Statistical Analysis 1: Comparison: Balanced Salt Solution (BSS) vs OMS302 Solution; Test type: Superiority or Other; p = 0.220, Wilcoxon rank-sum test — Treatment comparisons between OMS302 and each of the other three groups are based on Wilcoxon rank-sum test
Statistical Analysis 2: Comparison: OMS302 Mydriatic Solution (PE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.903, Wilcoxon rank-sum test — Treatment comparisons between OMS302 and each of the other three groups are based on Wilcoxon rank-sum test
Statistical Analysis 3: Comparison: OMS302 Anti-inflammatory Solution (KE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.463, Wilcoxon rank-sum test — Treatment comparisons between OMS302 and each of the other three groups are based on Wilcoxon rank-sum test

50. Secondary Outcome: Best Corrected Visual Acuity (BVCA) - Log Score, Day 30
Description: as for outcome 46
Time Frame: 30 days
Population: Subjects with scores at time point.
Measure: Mean (Standard Deviation); unit: Log score
Arm/Group | Balanced Salt Solution (BSS) | OMS302 Mydriatic Solution (PE) | OMS302 Anti-inflammatory Solution (KE) | OMS302 Solution
Number analyzed (Participants) | 56 | 55 | 55 | 54
Log score | 0.1 (0.2) | 0.1 (0.2) | 0.1 (0.2) | 0.1 (0.1)
Statistical Analysis 1: Comparison: Balanced Salt Solution (BSS) vs OMS302 Solution; Test type: Superiority or Other; p = 0.675, Wilcoxon rank-sum test — Treatment comparisons between OMS302 and each of the other three groups are based on Wilcoxon rank-sum test
Statistical Analysis 2: Comparison: OMS302 Mydriatic Solution (PE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.825, WIlcoxon rank-sum test — Treatment comparisons between OMS302 and each of the other three groups are based on Wilcoxon rank-sum test
Statistical Analysis 3: Comparison: OMS302 Anti-inflammatory Solution (KE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.668, Wilcoxon rank-sum test — Treatment comparisons between OMS302 and each of the other three groups are based on Wilcoxon rank-sum test

51. Secondary Outcome: Postoperative Ocular Inflammation in Summed Ocular Inflammation Score (SOIS) Grade, Baseline
Description: Postoperative inflammation as measured using the Summed Ocular Inflammation Score (SOIS), summarized by treatment arm and time point. Ocular inflammation was evaluated by measuring the anterior chamber cell count and flare using a slit lamp biomicroscope. SOIS was calculated by adding the average of subject's anterior chamber cells and flare grades. The minimum SOIS was 0 (indicating absence of inflammation), whereas the maximum SOIS was 8.
  Grading was as follows:
  Anterior Chamber Cells: Grade None = 0/no cells; Grade Mild = +1/1-5 cells; Grade Moderate = +2/6-15 cells; Grade Severe = +3/16-30 cells; Grade Very Severe = +4/>30 cells.
  Anterior Chamber Flare: Grade None = 0/no Tyndall effect; Grade Mild = +1/barely discernable Tyndall effect; Grade Moderate = +2/moderately intense Tyndall beam in anterior chamber; Grade Severe = +3/severely intense Tyndall beam; Grade Very Severe = +4/very severely intense Tyndall beam with a white and milky appearance to the aqueous
Time Frame: Baseline
Population: Subjects with scores at time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Balanced Salt Solution (BSS) | OMS302 Mydriatic Solution (PE) | OMS302 Anti-inflammatory Solution (KE) | OMS302 Solution
Number analyzed (Participants) | 56 | 56 | 55 | 55
units on a scale | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.1) | 0.0 (0.1)
Statistical Analysis 1: Comparison: Balanced Salt Solution (BSS) vs OMS302 Solution; Test type: Superiority or Other; p = 0.2066, ANOVA — Treatment comparisons between OMS302 and each of the other three groups are based on ANOVA model with covariates treatment group and the LOCS II grade group
Statistical Analysis 2: Comparison: OMS302 Mydriatic Solution (PE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.2066, ANOVA — [p-value comment as in outcome 51, analysis 1]
Statistical Analysis 3: Comparison: OMS302 Anti-inflammatory Solution (KE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.5263, ANOVA — [p-value comment as in outcome 51, analysis 1]

52. Secondary Outcome: Postoperative Ocular Inflammation in Summed Ocular Inflammation Score (SOIS) Grade, 2 Hours Post Surgery
Description: TPostoperative inflammation as measured using the Summed Ocular Inflammation Score (SOIS), summarized by treatment arm and time point. Ocular inflammation was evaluated by measuring the anterior chamber cell count and flare using a slit lamp biomicroscope. SOIS was calculated by adding the average of subject's anterior chamber cells and flare grades. The minimum SOIS was 0 (indicating absence of inflammation), whereas the maximum SOIS was 8.
  Grading was as follows:
  Anterior Chamber Cells: Grade None = 0/no cells; Grade Mild = +1/1-5 cells; Grade Moderate = +2/6-15 cells; Grade Severe = +3/16-30 cells; Grade Very Severe = +4/>30 cells.
  Anterior Chamber Flare: Grade None = 0/no Tyndall effect; Grade Mild = +1/barely discernable Tyndall effect; Grade Moderate = +2/moderately intense Tyndall beam in anterior chamber; Grade Severe = +3/severely intense Tyndall beam; Grade Very Severe = +4/very severely intense Tyndall beam with a white and milky appearance to the aqueous
Time Frame: Two hours
Population: Subjects with scores at time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Balanced Salt Solution (BSS) | OMS302 Mydriatic Solution (PE) | OMS302 Anti-inflammatory Solution (KE) | OMS302 Solution
Number analyzed (Participants) | 56 | 56 | 55 | 55
units on a scale | 2.7 (1.4) | 2.2 (1.3) | 2.5 (1.3) | 2.5 (1.2)
Statistical Analysis 1: Comparison: Balanced Salt Solution (BSS) vs OMS302 Solution; Test type: Superiority or Other; p = 0.4222, ANOVA — [p-value comment as in outcome 51, analysis 1]
Statistical Analysis 2: Comparison: OMS302 Mydriatic Solution (PE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.2712, ANOVA — [p-value comment as in outcome 51, analysis 1]
Statistical Analysis 3: Comparison: OMS302 Anti-inflammatory Solution (KE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.8819, ANOVA — [p-value comment as in outcome 51, analysis 1]

53. Secondary Outcome: Postoperative Ocular Inflammation in Summed Ocular Inflammation Score (SOIS) Grade, Day 1
Description: as for outcome 51
Time Frame: One day
Population: Subjects with scores at time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Balanced Salt Solution (BSS) | OMS302 Mydriatic Solution (PE) | OMS302 Anti-inflammatory Solution (KE) | OMS302 Solution
Number analyzed (Participants) | 56 | 56 | 55 | 55
units on a scale | 2.7 (1.4) | 2.3 (1.3) | 2.6 (1.3) | 2.2 (1.1)
Statistical Analysis 1: Comparison: Balanced Salt Solution (BSS) vs OMS302 Solution; Test type: Superiority or Other; p = 0.0510, ANOVA — [p-value comment as in outcome 51, analysis 1]
Statistical Analysis 2: Comparison: OMS302 Mydriatic Solution (PE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.8084, ANOVA — [p-value comment as in outcome 51, analysis 1]
Statistical Analysis 3: Comparison: OMS302 Anti-inflammatory Solution (KE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.1495, ANOVA — [p-value comment as in outcome 51, analysis 1]

54. Secondary Outcome: Postoperative Ocular Inflammation in Summed Ocular Inflammation Score (SOIS) Grade, Day 2
Description: as for outcome 51
Time Frame: Two days
Population: Subjects with scores at time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Balanced Salt Solution (BSS) | OMS302 Mydriatic Solution (PE) | OMS302 Anti-inflammatory Solution (KE) | OMS302 Solution
Number analyzed (Participants) | 56 | 56 | 55 | 55
units on a scale | 2.4 (1.3) | 2.0 (1.2) | 2.6 (1.4) | 2.2 (1.2)
Statistical Analysis 1: Comparison: Balanced Salt Solution (BSS) vs OMS302 Solution; Test type: Superiority or Other; p = 0.4099, ANOVA — [p-value comment as in outcome 51, analysis 1]
Statistical Analysis 2: Comparison: OMS302 Mydriatic Solution (PE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.6499, ANOVA — [p-value comment as in outcome 51, analysis 1]
Statistical Analysis 3: Comparison: OMS302 Anti-inflammatory Solution (KE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.0765, ANOVA — [p-value comment as in outcome 51, analysis 1]

55. Secondary Outcome: Postoperative Ocular Inflammation in Summed Ocular Inflammation Score (SOIS) Grade, Day 7
Description: as for outcome 51
Time Frame: Seven days
Population: Subjects with scores at time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Balanced Salt Solution (BSS) | OMS302 Mydriatic Solution (PE) | OMS302 Anti-inflammatory Solution (KE) | OMS302 Solution
Number analyzed (Participants) | 56 | 56 | 53 | 55
units on a scale | 1.5 (1.2) | 1.4 (1.2) | 1.5 (1.3) | 1.9 (1.3)
Statistical Analysis 1: Comparison: Balanced Salt Solution (BSS) vs OMS302 Solution; Test type: Superiority or Other; p = 0.0688, ANOVA — [p-value comment as in outcome 51, analysis 1]
Statistical Analysis 2: Comparison: OMS302 Mydriatic Solution (PE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.0314, ANOVA — [p-value comment as in outcome 51, analysis 1]
Statistical Analysis 3: Comparison: OMS302 Anti-inflammatory Solution (KE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.0775, ANOVA — [p-value comment as in outcome 51, analysis 1]

56. Secondary Outcome: Postoperative Ocular Inflammation in Summed Ocular Inflammation Score (SOIS) Grade, Day 14
Description: as for outcome 51
Time Frame: 14 days
Population: Subjects with scores at time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Balanced Salt Solution (BSS) | OMS302 Mydriatic Solution (PE) | OMS302 Anti-inflammatory Solution (KE) | OMS302 Solution
Number analyzed (Participants) | 55 | 56 | 55 | 53
units on a scale | 0.7 (0.7) | 0.6 (0.8) | 0.7 (0.9) | 0.8 (0.9)
Statistical Analysis 1: Comparison: Balanced Salt Solution (BSS) vs OMS302 Solution; Test type: Superiority or Other; p = 0.5369, ANOVA — [p-value comment as in outcome 51, analysis 1]
Statistical Analysis 2: Comparison: OMS302 Mydriatic Solution (PE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.3763, ANOVA — [p-value comment as in outcome 51, analysis 1]
Statistical Analysis 3: Comparison: OMS302 Anti-inflammatory Solution (KE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.6144, ANOVA — [p-value comment as in outcome 51, analysis 1]

57. Secondary Outcome: Postoperative Ocular Inflammation in Summed Ocular Inflammation Score (SOIS) Grade, Day 30
Description: as for outcome 51
Time Frame: 30 days
Population: Subjects with scores at time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Balanced Salt Solution (BSS) | OMS302 Mydriatic Solution (PE) | OMS302 Anti-inflammatory Solution (KE) | OMS302 Solution
Number analyzed (Participants) | 56 | 55 | 55 | 54
units on a scale | 0.4 (0.7) | 0.2 (0.5) | 0.3 (0.6) | 0.2 (0.4)
Statistical Analysis 1: Comparison: Balanced Salt Solution (BSS) vs OMS302 Solution; Test type: Superiority or Other; p = 0.1374, ANOVA — [p-value comment as in outcome 51, analysis 1]
Statistical Analysis 2: Comparison: OMS302 Mydriatic Solution (PE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.9146, ANOVA — [p-value comment as in outcome 51, analysis 1]
Statistical Analysis 3: Comparison: OMS302 Anti-inflammatory Solution (KE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.7599, ANOVA — [p-value comment as in outcome 51, analysis 1]

58. Secondary Outcome: Subjects With Postoperative Ocular Inflammation SOIS = 0, Baseline
Description: Number of subjects with Summed Ocular Inflammation Score (SOIS) = 0, summarized by treatment arm and time point. Ocular inflammation was evaluated by measuring the anterior chamber cell count and flare using a slit lamp biomicroscope. SOIS was calculated by adding the average of subject's anterior chamber cells and flare grades. The minimum SOIS was 0 (indicating absence of inflammation), whereas the maximum SOIS was 8.
  Grading was as follows:
  Anterior Chamber Cells: Grade None = 0/no cells; Grade Mild = +1/1-5 cells; Grade Moderate = +2/6-15 cells; Grade Severe = +3/16-30 cells; Grade Very Severe = +4/>30 cells.
  Anterior Chamber Flare: Grade None = 0/no Tyndall effect; Grade Mild = +1/barely discernable Tyndall effect; Grade Moderate = +2/moderately intense Tyndall beam in anterior chamber; Grade Severe = +3/severely intense Tyndall beam; Grade Very Severe = +4/very severely intense Tyndall beam with a white and milky appearance to the aqueous
Time Frame: Baseline
Population: Subjects with scores at time point.
Measure: Number; unit: participants
Arm/Group | Balanced Salt Solution (BSS) | OMS302 Mydriatic Solution (PE) | OMS302 Anti-inflammatory Solution (KE) | OMS302 Solution
Number analyzed (Participants) | 56 | 56 | 55 | 55
participants | 56 | 56 | 54 | 54
Statistical Analysis 1: Comparison: Balanced Salt Solution (BSS) vs OMS302 Solution; Test type: Superiority or Other; p = 0.317, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]
Statistical Analysis 2: Comparison: OMS302 Mydriatic Solution (PE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.317, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]
Statistical Analysis 3: Comparison: OMS302 Anti-inflammatory Solution (KE) vs OMS302 Solution; Test type: Superiority or Other; p = 1.000, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]

59. Secondary Outcome: Subjects With Postoperative Ocular Inflammation SOIS = 0, Two Hours Post-surgery
Description: as for outcome 58
Time Frame: Two hours
Population: Subjects with scores at time point.
Measure: Number; unit: participants
Arm/Group | Balanced Salt Solution (BSS) | OMS302 Mydriatic Solution (PE) | OMS302 Anti-inflammatory Solution (KE) | OMS302 Solution
Number analyzed (Participants) | 56 | 56 | 55 | 55
participants | 1 | 3 | 1 | 2
Statistical Analysis 1: Comparison: Balanced Salt Solution (BSS) vs OMS302 Solution; Test type: Superiority or Other; p = 0.559, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]
Statistical Analysis 2: Comparison: OMS302 Mydriatic Solution (PE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.647, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]
Statistical Analysis 3: Comparison: OMS302 Anti-inflammatory Solution (KE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.559, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]

60. Secondary Outcome: Subjects With Postoperative Ocular Inflammation SOIS = 0, Day 1
Description: as for outcome 58
Time Frame: One day
Population: Subjects with scores at time point.
Measure: Number; unit: participants
Arm/Group | Balanced Salt Solution (BSS) | OMS302 Mydriatic Solution (PE) | OMS302 Anti-inflammatory Solution (KE) | OMS302 Solution
Number analyzed (Participants) | 56 | 56 | 55 | 55
participants | 1 | 1 | 1 | 0
Statistical Analysis 1: Comparison: Balanced Salt Solution (BSS) vs OMS302 Solution; Test type: Superiority or Other; p = 0.317, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]
Statistical Analysis 2: Comparison: OMS302 Mydriatic Solution (PE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.335, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]
Statistical Analysis 3: Comparison: OMS302 Anti-inflammatory Solution (KE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.317, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]

61. Secondary Outcome: Subjects With Postoperative Ocular Inflammation SOIS = 0, Day 2
Description: as for outcome 58
Time Frame: Two days
Population: Subjects with scores at time point.
Measure: Number; unit: participants
Arm/Group | Balanced Salt Solution (BSS) | OMS302 Mydriatic Solution (PE) | OMS302 Anti-inflammatory Solution (KE) | OMS302 Solution
Number analyzed (Participants) | 56 | 56 | 55 | 55
participants | 1 | 2 | 1 | 1
Statistical Analysis 1: Comparison: Balanced Salt Solution (BSS) vs OMS302 Solution; Test type: Superiority or Other; p = 1.000, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]
Statistical Analysis 2: Comparison: OMS302 Mydriatic Solution (PE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.559, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]
Statistical Analysis 3: Comparison: OMS302 Anti-inflammatory Solution (KE) vs OMS302 Solution; Test type: Superiority or Other; p = 1.000, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]

62. Secondary Outcome: Subjects With Postoperative Ocular Inflammation SOIS = 0, Day 7
Description: as for outcome 58
Time Frame: Seven days
Population: Subjects with scores at time point.
Measure: Number; unit: participants
Arm/Group | Balanced Salt Solution (BSS) | OMS302 Mydriatic Solution (PE) | OMS302 Anti-inflammatory Solution (KE) | OMS302 Solution
Number analyzed (Participants) | 56 | 56 | 53 | 55
participants | 9 | 11 | 12 | 8
Statistical Analysis 1: Comparison: Balanced Salt Solution (BSS) vs OMS302 Solution; Test type: Superiority or Other; p = 0.824, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]
Statistical Analysis 2: Comparison: OMS302 Mydriatic Solution (PE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.476, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]
Statistical Analysis 3: Comparison: OMS302 Anti-inflammatory Solution (KE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.281, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]

63. Secondary Outcome: Subjects With Postoperative Ocular Inflammation SOIS = 0, Day 14
Description: as for outcome 58
Time Frame: 14 days
Population: Subjects with scores at time point.
Measure: Number; unit: participants
Arm/Group | Balanced Salt Solution (BSS) | OMS302 Mydriatic Solution (PE) | OMS302 Anti-inflammatory Solution (KE) | OMS302 Solution
Number analyzed (Participants) | 55 | 56 | 55 | 53
participants | 25 | 29 | 28 | 25
Statistical Analysis 1: Comparison: Balanced Salt Solution (BSS) vs OMS302 Solution; Test type: Superiority or Other; p = 0.842, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]
Statistical Analysis 2: Comparison: OMS302 Mydriatic Solution (PE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.619, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]
Statistical Analysis 3: Comparison: OMS302 Anti-inflammatory Solution (KE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.711, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]

64. Secondary Outcome: Subjects With Postoperative Ocular Inflammation SOIS = 0, Day 30
Description: as for outcome 58
Time Frame: 30 days
Population: Subjects with scores at time point.
Measure: Number; unit: participants
Arm/Group | Balanced Salt Solution (BSS) | OMS302 Mydriatic Solution (PE) | OMS302 Anti-inflammatory Solution (KE) | OMS302 Solution
Number analyzed (Participants) | 56 | 55 | 55 | 54
participants | 40 | 43 | 42 | 40
Statistical Analysis 1: Comparison: Balanced Salt Solution (BSS) vs OMS302 Solution; Test type: Superiority or Other; p = 0.773, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]
Statistical Analysis 2: Comparison: OMS302 Mydriatic Solution (PE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.592, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]
Statistical Analysis 3: Comparison: OMS302 Anti-inflammatory Solution (KE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.787, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]

65. Secondary Outcome: Postoperative Mean Anterior Chamber Cell Count, Two Hours Post-Surgery
Description: The mean anterior chamber cell count was calculated as the average of the two anterior chamber cell counts. If a cell count was indicated as > 30, it was imputed as 45 for the purpose of treatment comparisons which was performed using pairwise Wilcoxon tests.
Time Frame: Two hours
Population: Subjects with data at time point.
Measure: Mean (Standard Deviation); unit: cells
Arm/Group | Balanced Salt Solution (BSS) | OMS302 Mydriatic Solution (PE) | OMS302 Anti-inflammatory Solution (KE) | OMS302 Solution
Number analyzed (Participants) | 54 | 52 | 53 | 53
cells | 11.2 (9.4) | 9.2 (11.1) | 10.9 (10.1) | 10.3 (8.6)
Statistical Analysis 1: Comparison: Balanced Salt Solution (BSS) vs OMS302 Solution; Test type: Superiority or Other; p = 0.695, Wilcoxon rank-sum test — Treatment comparisons between OMS302 and each of the other three groups were based on Wilcoxon rank-sum test. For subjects with mean count > 30, the mean count was imputed as 45 for the purpose of treatment comparisons
Statistical Analysis 2: Comparison: OMS302 Mydriatic Solution (PE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.166, Wilcoxon rank-sum test — [p-value comment as in outcome 65, analysis 1]
Statistical Analysis 3: Comparison: OMS302 Anti-inflammatory Solution (KE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.987, Wilcoxon rank-sum test — [p-value comment as in outcome 65, analysis 1]

66. Secondary Outcome: Postoperative Mean Anterior Chamber Cell Count, Day 1
Description: as for outcome 65
Time Frame: One day
Population: Subjects with data at time point.
Measure: Mean (Standard Deviation); unit: cells
Arm/Group | Balanced Salt Solution (BSS) | OMS302 Mydriatic Solution (PE) | OMS302 Anti-inflammatory Solution (KE) | OMS302 Solution
Number analyzed (Participants) | 53 | 55 | 54 | 53
cells | 11.2 (9.5) | 9.3 (9.7) | 10.4 (8.9) | 8.4 (6.7)
Statistical Analysis 1: Comparison: Balanced Salt Solution (BSS) vs OMS302 Solution; Test type: Superiority or Other; p = 0.134, Wilcoxon rank-sum test — [p-value comment as in outcome 65, analysis 1]
Statistical Analysis 2: Comparison: OMS302 Mydriatic Solution (PE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.710, Wilcoxon rank-sum test — [p-value comment as in outcome 65, analysis 1]
Statistical Analysis 3: Comparison: OMS302 Anti-inflammatory Solution (KE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.310, Wilcoxon rank-sum test — [p-value comment as in outcome 65, analysis 1]

67. Secondary Outcome: Postoperative Mean Anterior Chamber Cell Count, Day 2
Description: as for outcome 65
Time Frame: Two days
Population: Subjects with data at time point.
Measure: Mean (Standard Deviation); unit: cells
Arm/Group | Balanced Salt Solution (BSS) | OMS302 Mydriatic Solution (PE) | OMS302 Anti-inflammatory Solution (KE) | OMS302 Solution
Number analyzed (Participants) | 54 | 54 | 53 | 54
cells | 9.1 (6.4) | 6.8 (7.8) | 10.2 (7.6) | 7.2 (6.0)
Statistical Analysis 1: Comparison: Balanced Salt Solution (BSS) vs OMS302 Solution; Test type: Superiority or Other; p = 0.086, Wilcoxon rank-sum test — [p-value comment as in outcome 65, analysis 1]
Statistical Analysis 2: Comparison: OMS302 Mydriatic Solution (PE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.183, Wilcoxon rank-sum test — [p-value comment as in outcome 65, analysis 1]
Statistical Analysis 3: Comparison: OMS302 Anti-inflammatory Solution (KE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.029, Wilcoxon rank-sum test — [p-value comment as in outcome 65, analysis 1]

68. Secondary Outcome: Postoperative Mean Anterior Chamber Cell Count, Day 7
Description: as for outcome 65
Time Frame: Seven days
Population: Subjects with data at time point.
Measure: Mean (Standard Deviation); unit: cells
Arm/Group | Balanced Salt Solution (BSS) | OMS302 Mydriatic Solution (PE) | OMS302 Anti-inflammatory Solution (KE) | OMS302 Solution
Number analyzed (Participants) | 55 | 55 | 52 | 54
cells | 4.5 (5.2) | 4.2 (7.5) | 3.6 (4.6) | 6.9 (10.1)
Statistical Analysis 1: Comparison: Balanced Salt Solution (BSS) vs OMS302 Solution; Test type: Superiority or Other; p = 0.206, Wilcoxon rank-sum test — [p-value comment as in outcome 65, analysis 1]
Statistical Analysis 2: Comparison: OMS302 Mydriatic Solution (PE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.021, Wilcoxon rank-sum test — [p-value comment as in outcome 65, analysis 1]
Statistical Analysis 3: Comparison: OMS302 Anti-inflammatory Solution (KE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.026, Wilcoxon rank-sum test — [p-value comment as in outcome 65, analysis 1]

69. Secondary Outcome: Postoperative Mean Anterior Chamber Cell Count, Day 14
Description: as for outcome 65
Time Frame: 14 days
Population: Subjects with data at time point.
Measure: Mean (Standard Deviation); unit: cells
Arm/Group | Balanced Salt Solution (BSS) | OMS302 Mydriatic Solution (PE) | OMS302 Anti-inflammatory Solution (KE) | OMS302 Solution
Number analyzed (Participants) | 54 | 55 | 54 | 52
cells | 1.6 (2.1) | 1.3 (2.4) | 1.6 (2.7) | 2.1 (3.9)
Statistical Analysis 1: Comparison: Balanced Salt Solution (BSS) vs OMS302 Solution; Test type: Superiority or Other; p = 0.822, Wilcoxon rank-sum test — [p-value comment as in outcome 65, analysis 1]
Statistical Analysis 2: Comparison: OMS302 Mydriatic Solution (PE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.424, Wilcoxon rank-sum test — [p-value comment as in outcome 65, analysis 1]
Statistical Analysis 3: Comparison: OMS302 Anti-inflammatory Solution (KE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.695, Wilcoxon rank-sum test — [p-value comment as in outcome 65, analysis 1]

70. Secondary Outcome: Postoperative Mean Anterior Chamber Cell Count, Day 30
Description: as for outcome 65
Time Frame: 30 days
Population: Subjects with data at time point.
Measure: Mean (Standard Deviation); unit: cells
Arm/Group | Balanced Salt Solution (BSS) | OMS302 Mydriatic Solution (PE) | OMS302 Anti-inflammatory Solution (KE) | OMS302 Solution
Number analyzed (Participants) | 55 | 55 | 55 | 53
cells | 1.1 (2.3) | 0.3 (0.8) | 0.5 (1.2) | 0.5 (1.2)
Statistical Analysis 1: Comparison: Balanced Salt Solution (BSS) vs OMS302 Solution; Test type: Superiority or Other; p = 0.489, Wilcoxon rank-sum test — [p-value comment as in outcome 65, analysis 1]
Statistical Analysis 2: Comparison: OMS302 Mydriatic Solution (PE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.459, Wilcoxon rank-sum test — [p-value comment as in outcome 65, analysis 1]
Statistical Analysis 3: Comparison: OMS302 Anti-inflammatory Solution (KE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.990, Wilcoxon rank-sum test — [p-value comment as in outcome 65, analysis 1]

71. Secondary Outcome: Ocular Pain VAS Score After Day 0
Description: VAS pain scores (where 0 = no pain and 100 = worst possible pain) after the day of surgery were summarized.
Time Frame: 43 days
Population: Subjects with data at time point.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Balanced Salt Solution (BSS) | OMS302 Mydriatic Solution (PE) | OMS302 Anti-inflammatory Solution (KE) | OMS302 Solution
Number analyzed (Participants) | 56 | 56 | 55 | 55
mm
  Day 1 AM; n = 55, 54, 55, 55 | 13.4 (21.7) | 13.0 (18.1) | 2.7 (8.3) | 7.7 (18.4)
  Day 1 PM; n = 54, 54, 51, 51 | 6.6 (10.2) | 12.6 (19.4) | 6.8 (15.1) | 11.6 (20.6)
  Day 2 AM; n = 55, 55, 55, 54 | 7.7 (11.1) | 10.8 (18.2) | 9.5 (18.9) | 10.9 (13.7)
  Day 2 PM; n = 52, 55, 53, 53 | 5.3 (9.4) | 7.3 (15.5) | 7.2 (15.4) | 6.4 (11.8)
  Day 3 AM; n = 53, 53, 53, 49 | 4.1 (7.0) | 5.4 (11.5) | 4.8 (11.3) | 8.9 (18.8)
  Day 3 PM; n = 53, 55, 55, 50 | 4.7 (9.8) | 5.1 (11.0) | 3.7 (8.7) | 4.4 (10.7)
  Day 4 AM; n = 52, 53, 52, 48 | 2.8 (6.0) | 3.5 (8.3) | 3.9 (10.8) | 5.0 (10.5)
  Day 4 PM; n = 53, 52, 55, 52 | 4.5 (9.2) | 3.7 (9.4) | 4.8 (14.2) | 4.1 (8.3)
  Day 5 AM; n = 54, 54, 53, 50 | 3.6 (9.9) | 6.4 (18.5) | 3.4 (10.6) | 6.5 (14.8)
  Day 5 PM; n = 54, 55, 54, 51 | 3.9 (8.5) | 3.9 (10.4) | 3.3 (9.6) | 5.2 (12.5)
  Day 6 AM; n = 53, 54, 53, 50 | 3.5 (6.3) | 4.6 (13.3) | 3.6 (10.2) | 6.0 (14.3)
  Day 6 PM; n = 54, 53, 54, 50 | 2.9 (5.5) | 4.0 (11.0) | 2.7 (9.3) | 4.6 (12.2)
  Day 7; n = 54, 54, 54, 53 | 2.1 (5.3) | 3.5 (9.0) | 3.3 (11.0) | 4.5 (13.9)
  Day 8; n = 22, 28, 21, 13 | 1.3 (2.3) | 4.9 (14.7) | 0.6 (1.0) | 2.2 (6.3)
  Day 9; n = 4, 4, 3, 2 | 0.0 (0.0) | 0.3 (0.5) | 0.0 (0.0) | 0.0 (0.0)
  Day 10; 1, 2, 3, 1 | 0.0 (0) | 0.5 (0.7) | 0.0 (0.0) | 0.0 (0)
  Day 11; n = 1, 2, 4, 1 | 0.0 (0) | 0.5 (0.7) | 0.0 (0.0) | 0.0 (0)
  Day 12; n = 2, 2, 2, 1 | 2.5 (3.5) | 0.5 (0.7) | 0.0 (0.0) | 0.0 (0)
  Day 13; n = 11, 8, 15, 9 | 1.1 (3.3) | 0.3 (0.5) | 0.7 (1.8) | 0.0 (0.0)
  Day 14; n = 17, 16, 21, 26 | 2.7 (7.7) | 0.2 (0.5) | 1.0 (2.2) | 0.6 (1.4)
  Day 15; 22, 25, 18, 14 | 2.1 (3.6) | 1.8 (8.0) | 0.2 (0.4) | 4.5 (13.4)
  Day 16; 1, 7, 2, 5 | 0.0 (0) | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0)
  Day 17; n = 2, 0, 0, 1 | 4.5 (6.4) | NA (NA) — Subjects not available for assessment at time point | NA (NA) — Subjects not available for assessment at time point | 0.0 (0)
  Day 18; n = 0, 0, 1, 0 | NA (NA) — Subjects not available for assessment at time point | NA (NA) — Subjects not available for assessment at time point | 0.0 (0) | NA (NA) — Subjects not available for assessment at time point
  Day 19; n = 1, 0, 0, 0 | 0.0 (0) | NA (NA) — Subjects not available for assessment at time point | NA (NA) — Subjects not available for assessment at time point | NA (NA) — Subjects not available for assessment at time point
  Day 20; n = 0, 1, 0, 0 | NA (NA) — Subjects not available for assessment at time point | 0.0 (0) | NA (NA) — Subjects not available for assessment at time point | NA (NA) — Subjects not available for assessment at time point
  Day 21; n = 1, 0, 0, 0 | 0.0 (0) | NA (NA) — Subjects not available for assessment at time point | NA (NA) — Subjects not available for assessment at time point | NA (NA) — Subjects not available for assessment at time point
  Day 22; n = 0, 1, 1, 0 | NA (NA) — Subjects not available for assessment at time point | 0.0 (0) | 0.0 (0) | NA (NA) — Subjects not available for assessment at time point
  Day 26; n = 0, 1, 0, 0 | NA (NA) — Subjects not available for assessment at time point | 0.0 (0) | NA (NA) — Subjects not available for assessment at time point | NA (NA) — Subjects not available for assessment at time point
  Day 27; n = 9, 9, 6, 5 | 0.6 (1.7) | 0.1 (0.3) | 0.0 (0.0) | 0.2 (0.4)
  Day 28; n = 11, 12, 14, 25 | 0.6 (0.9) | 0.0 (0.0) | 0.8 (2.2) | 0.2 (0.7)
  Day 29; n = 16, 14, 18, 13 | 0.1 (0.3) | 0.1 (0.3) | 1.6 (5.1) | 0.0 (0.0)
  Day 30; n = 15, 13, 6, 5 | 0.8 (2.8) | 0.3 (0.9) | 0.0 (0.0) | 0.8 (1.8)
  Day 31; n = 2, 2, 1, 3 | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0) | 0.0 (0.0)
  Day 32; n = 0, 0, 5, 0 | NA (NA) — Subjects not available for assessment at time point | NA (NA) — Subjects not available for assessment at time point | 0.0 (0.0) | NA (NA) — Subjects not available for assessment at time point
  Day 33;n = 0, 0, 2, 0 | NA (NA) — Subjects not available for assessment at time point | NA (NA) — Subjects not available for assessment at time point | 0.0 (0.0) | NA (NA) — Subjects not available for assessment at time point
  Day 34; n = 1, 0, 0, 0 | 0.0 (0) | NA (NA) — Subjects not available for assessment at time point | NA (NA) — Subjects not available for assessment at time point | NA (NA) — Subjects not available for assessment at time point
  Day 35; n = 1, 0, 1, 1 | 0.0 (0) | NA (NA) — Subjects not available for assessment at time point | 0.0 (0) | 0.0 (0)
  Day 36; n = 1, 1, 1, 1 | 0.0 (0) | 50.0 (0) | 0.0 (0) | 0.0 (0)
  Day 37; n = 0, 1, 0, 0 | NA (NA) — Subjects not available for assessment at time point | 0.0 (0) | NA (NA) — Subjects not available for assessment at time point | NA (NA) — Subjects not available for assessment at time point
  Day 43; n = 0, 1, 0, 0 | NA (NA) — Subjects not available for assessment at time point | 0.0 (0) | NA (NA) — Subjects not available for assessment at time point | NA (NA) — Subjects not available for assessment at time point

72. Secondary Outcome: Postoperative Use of Ophthalmic Anti-inflammatory Medications
Description: Ophthalmic anti-inflammatory medications were identified by reviewing concomitant medications. Subject incidence of ophthalmic anti-inflammatory medication use by post-surgery day was presented. Treatment comparisons were performed using a Cochran-Mantel- Haenszel (CMH) test adjusting for the stratification factor LOCS II grade.
Time Frame: up to 30 days
Population: All randomized subjects
Measure: Number; unit: participants
Arm/Group | Balanced Salt Solution (BSS) | OMS302 Mydriatic Solution (PE) | OMS302 Anti-inflammatory Solution (KE) | OMS302 Solution
Number analyzed (Participants) | 56 | 56 | 55 | 56
participants
  Bromfenac sodium | 2 | 9 | 8 | 6
  Dexamethasone | 1 | 0 | 0 | 2
  Difluprednate | 6 | 8 | 7 | 7
  Ketorlac | 0 | 0 | 1 | 0
  Ketorolac tromethamine | 0 | 1 | 0 | 0
  Loteprednol etabonate | 0 | 1 | 1 | 0
  Nepafenac | 10 | 4 | 7 | 4
  Prednisolone acetate | 25 | 29 | 28 | 29
Statistical Analysis 1: Comparison: Balanced Salt Solution (BSS) vs OMS302 Solution; Test type: Superiority or Other; p = 0.4575, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]
Statistical Analysis 2: Comparison: OMS302 Mydriatic Solution (PE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.8318, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]
Statistical Analysis 3: Comparison: OMS302 Anti-inflammatory Solution (KE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.8946, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]

73. Secondary Outcome: Use of Pain Medications at Day 1
Description: Ocular pain medications were identified by reviewing concomitant medications. Subject incidence of ocular pain medication use at day 1 and post day 1 were presented. Treatment comparisons were performed using a Cochran-Mantel- Haenszel (CMH) test adjusting for the stratification factor LOCS II grade.
Time Frame: One day
Population: All randomized subjects
Measure: Number; unit: participants
Arm/Group | Balanced Salt Solution (BSS) | OMS302 Mydriatic Solution (PE) | OMS302 Anti-inflammatory Solution (KE) | OMS302 Solution
Number analyzed (Participants) | 56 | 56 | 55 | 56
participants
  Axotal | 0 | 0 | 0 | 1
  Diclofenac | 1 | 0 | 0 | 0
  Ibuprofen | 1 | 0 | 1 | 0
  Naproxen Sodium | 0 | 0 | 1 | 0
  Paracetamol | 23 | 26 | 9 | 18
  Tramadol | 0 | 2 | 0 | 0
Statistical Analysis 1: Comparison: Balanced Salt Solution (BSS) vs OMS302 Solution; Test type: Superiority or Other; p = 0.1570, Cochran-Mantel-Haenszel — Ocular pain medications will be identified by reviewing concomitant medications. Subject incidence of ocular pain medication use at day 1 and post day 1 will be presented. Treatment comparisons will be performed using methodology 1
Statistical Analysis 2: Comparison: OMS302 Mydriatic Solution (PE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.0839, Cochran-Mantel-Haenszel — [p-value comment as in outcome 73, analysis 1]
Statistical Analysis 3: Comparison: OMS302 Anti-inflammatory Solution (KE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.0920, Cochran-Mantel-Haenszel — [p-value comment as in outcome 73, analysis 1]

74. Secondary Outcome: Use of Pain Medications After Day 1
Description: as for outcome 73
Time Frame: up to 30 days
Population: All randomized subjects
Measure: Number; unit: participants
Arm/Group | Balanced Salt Solution (BSS) | OMS302 Mydriatic Solution (PE) | OMS302 Anti-inflammatory Solution (KE) | OMS302 Solution
Number analyzed (Participants) | 56 | 56 | 55 | 56
participants
  Axotal | 0 | 0 | 0 | 1
  Celecoxib | 1 | 0 | 0 | 0
  Diclofenac | 1 | 0 | 0 | 0
  Hydrocodone | 1 | 0 | 0 | 0
  Ibuprofen | 1 | 0 | 0 | 0
  Naproxen | 1 | 0 | 0 | 0
  Naproxen Sodium | 0 | 0 | 0 | 1
  Paracetamol | 23 | 21 | 20 | 29
  Tramadol | 0 | 2 | 0 | 0
  Tylox | 0 | 1 | 0 | 0
Statistical Analysis 1: Comparison: Balanced Salt Solution (BSS) vs OMS302 Solution; Test type: Superiority or Other; p = 0.711, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]
Statistical Analysis 2: Comparison: OMS302 Mydriatic Solution (PE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.253, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]
Statistical Analysis 3: Comparison: OMS302 Anti-inflammatory Solution (KE) vs OMS302 Solution; Test type: Superiority or Other; p = 0.104, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Balanced Salt Solution (BSS) | OMS302 Mydriatic Solution (PE) | OMS302 Anti-inflammatory Solution (KE) | OMS302 Solution
Serious Adverse Events (participants affected / at risk) | 0/57 | 1/54 | 0/55 | 0/56
Other Adverse Events (participants affected / at risk) | 45/57 | 43/54 | 37/55 | 47/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Balanced Salt Solution (BSS) (N=57) | OMS302 Mydriatic Solution (PE) (N=54) | OMS302 Anti-inflammatory Solution (KE) (N=55) | OMS302 Solution (N=56)
Facial neuralgia (Nervous system disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Balanced Salt Solution (BSS) (N=57) | OMS302 Mydriatic Solution (PE) (N=54) | OMS302 Anti-inflammatory Solution (KE) (N=55) | OMS302 Solution (N=56)
Eye pain (Eye disorders) | 16 | 21 | 13 | 17
Inflammation (General disorders) | 13 | 12 | 8 | 11
Eye inflammation (Eye disorders) | 5 | 9 | 12 | 11
Pain (General disorders) | 11 | 8 | 8 | 9
Headache (Nervous system disorders) | 5 | 2 | 4 | 4
Photophobia (Eye disorders) | 1 | 3 | 2 | 4
Iritis (Eye disorders) | 0 | 2 | 2 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI agreed not to publish or otherwise to disclose Study data without prior written consent from the sponsor for a period of 24 months following Study completion or until data are published in a combined publication (whichever occurs first). The sponsor can review communications containing results prior to public release and embargo those communications for a period that is no longer than 60 days from the date of receipt of the non-public communication. The sponsor cannot extend the embargo.